CLINICAL TRIAL: NCT00048581
Title: A Phase III, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of BMS-188667 in Subjects With Active Rheumatoid Arthritis on Background Disease Modifying Anti-Rheumatic Drugs (DMARDS) Who Have Failed Anti-Tumor Necrosis Factor (TNF) Therapy
Brief Title: Phase III Study of BMS-188667 (CTLA4Ig) in Patients With Rheumatoid Arthritis Who Are Currently Failing Anti-TNF Therapy or Who Have Failed Anti-TNF Therapy in the Past.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-029
Record Dates: First submitted 2002-11-02; First posted 2002-11-13 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Abatacept (Active Comparator): Short Term Portion of Study
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): Short Term Portion of Study
  Interventions: Drug: Placebo
- Abatacept (Long Term) (Active Comparator): Long Term Portion of Study:
  All participants receive Active Drug
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Vials, intravenous (IV), ~10mg/kg abatacept, One every 2 weeks for first month then every 4 weeks thereafter, 6 months.
  Other Names: Orencia; BMS-188667; CTLA4Ig
  Arms: Abatacept
Drug: Placebo — Vials, IV, 0mg, One every 2 weeks for first month then every 4 weeks thereafter, 6 months.
  Arms: Placebo
Drug: Abatacept — Vials, IV, ~10mg/kg abatacept, every 4 weeks, 5.5 years
  Other Names: Orencia; BMS-188667; CTLA4Ig
  Arms: Abatacept (Long Term)

SUMMARY:
The purpose of this clinical research study is to determine whether abatacept treatment on a background of Disease Modifying Antirheumatic Drugs (DMARDs) will relieve the symptoms of rheumatoid arthritis (RA) in participants who are currently receiving anti-tumor necrosis factor (TNF) therapy for at least 3 months and are not responding or have taken anti-TNF therapy in the last 3 months and did not respond. The safety of treatment with abatacept will also be evaluated. This study also has a 4.5-year long-term extension beginning 6 months after the start of the study.

ELIGIBILITY:
Eligibility Criteria:

* Active rheumatoid arthritis currently failing anti-TNF therapy or have failed anti-TNF therapy in the past.

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Current symptoms of serious medical disease
* History of cancer in last 5 years other than non-melanoma skin cancer
* Chronic serious infection
* Active TB requiring treatment in last 5 years
* Herpes zoster in last 2 months
* Any active viral infection including Human Immunodeficiency Virus (HIV)
* Serious side effects associated with previous anti-TNF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2002-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Paradise Valley, Arizona
  - Local Institution, La Jolla, California
  - Local Institution, Long Beach, California
  - Local Institution, Palo Alto, California
  - Local Institution, Rancho Mirage, California
  - Local Institution, Denver, Colorado
  - Local Institution, Englewood, Colorado
  - Local Institution, Bridgeport, Connecticut
  - Local Institution, Hamden, Connecticut
  - Local Institution, Clearwater, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Largo, Florida
  - Local Institution, Palm Harbor, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Rome, Georgia
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Wichita, Kansas
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Boston, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Lincoln, Nebraska
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Albany, New York
  - Local Institution, Syracuse, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Bismarck, North Dakota
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Eugene, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Duncansville, Pennsylvania
  - Local Institution, Norristown, Pennsylvania
  - Local Institution, Sellersville, Pennsylvania
  - Local Institution, Willow Grove, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Vancouver, Washington
  - Local Institution, Milwaukee, Wisconsin

REFERENCES:
- [Background] Hassett AL, Li T, Buyske S, Savage SV, Gignac MA. The multi-faceted assessment of independence in patients with rheumatoid arthritis: preliminary validation from the ATTAIN study. Curr Med Res Opin. 2008 May;24(5):1443-53. doi: 10.1185/030079908x297376. Epub 2008 Apr 9. PMID 18402714
- [Background] Stewart AL and Ware JE. Measuring function and well being. The Medical Outcomes Study Approach. Durham, NC: Duke University Press. 1992.
- [Background] Spritzer KL, Hays RD. (2003, November). MOS Sleep Scale: A Manual For Use and Scoring, Version 1.0. Los Angeles, CA.
- [Derived] Alten R, Burkhardt H, Feist E, Kruger K, Rech J, Rubbert-Roth A, Voll RE, Elbez Y, Rauch C. Abatacept used in combination with non-methotrexate disease-modifying antirheumatic drugs: a descriptive analysis of data from interventional trials and the real-world setting. Arthritis Res Ther. 2018 Jan 2;20(1):1. doi: 10.1186/s13075-017-1488-5. PMID 29329602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 738 participants were enrolled and 393 participants were randomized. Two participants were randomized in error and were not treated.
Groups:
- Abatacept (ABA): Participants with active RA who met the inclusion/exclusion criteria for this study were randomized to receive abatacept on a background of DMARDs. Participants must have been treated with anti-TNF therapy for at least 3 months and designated as anti-TNF therapy failures due to inadequate efficacy. Participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram. Study medication was administered on Days 1, 15, 29 and every 28 days thereafter for a total of 7 doses. Each dose was infused intravenously over approximately 30 minutes.
- Placebo (PLA): Participants with active RA who met the inclusion/exclusion criteria for this study were randomized to receive placebo on a background of DMARDs. Participants must have been treated with anti-TNF therapy for at least 3 months and designated as anti-TNF therapy failures due to inadequate efficacy. Placebo was administered IV on Days 1, 15, 29, 57, 85, 113, and 141.
- Open-label ABA: All participants who completed the double-blind period were eligible to continue in the open-label period. At the beginning of the open-label period (Day 169), all eligible participants were re-allocated to a 10 mg/kg weight-tiered dose of abatacept at their enrollment visit into the open-label period, based on their entry weight into the study. Participant dose was adjusted based on annual anniversary weight. Participants weighing > 100 kg received 1 g, participants weighing ≥ 60 kg and ≤ 100 kg received 750 mg, and participants weighing < 60 kg received 500 mg on a background of DMARDs (at discretion of the investigator). Concomitant biologic RA therapies were later excluded.
Period: Double-Blind Period
Arm/Group | Abatacept (ABA) | Placebo (PLA) | Open-label ABA
Started | 258 | 133 | 0
Completed | 223 | 99 | 0
Not Completed | 35 | 34 | 0
Not completed — Adverse Event | 9 | 5 | 0
Not completed — Lack of Efficacy | 14 | 27 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 0
Not completed — Participant Has History of Lymphopenia | 1 | 0 | 0
Not completed — Investigator Decision | 1 | 0 | 0
Period: Open-Label Period
Arm/Group | Abatacept (ABA) | Placebo (PLA) | Open-label ABA
Started | 0 | 0 | 317
Completed | 0 | 0 | 150
Not Completed | 0 | 0 | 167
Not completed — Death | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 37
Not completed — Lack of Efficacy | 0 | 0 | 69
Not completed — Lost to Follow-up | 0 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 20
Not completed — No Longer Meets Study Criteria | 0 | 0 | 2
Not completed — Poor/Non-compliance | 0 | 0 | 5
Not completed — Pregnancy | 0 | 0 | 7
Not completed — Study Site Closure | 0 | 0 | 2
Not completed — Continue ABA With Primary Rheumatologist | 0 | 0 | 3
Not completed — Problem With Transportation To Site | 0 | 0 | 1
Not completed — Primary Investigator Retired | 0 | 0 | 2
Not completed — Study Ended By Sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept (ABA) | Placebo (PLA) | Total
Number analyzed (Participants) | 258 | 133 | 391
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.4) | 52.7 (11.3) | 53.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 106 | 305
  Male | 59 | 27 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 248 | 124 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  North America | 189 | 99 | 288
  Europe | 69 | 34 | 103
Weight [Mean (Standard Deviation); unit: kg] | 78.2 (19.0) | 78.2 (21.0) | 78.2 (19.7)

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Period (DB); Number of Participants With American College of Rheumatology (ACR) 20 Response at Day 169
Description: ACR 20 response requires a participant to have a 20% reduction in the number of swollen and tender joints, and a reduction of 20% in three of the following five parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in Health Assessment Questionnaire (HAQ) score. A participant achieved a sustained ACR 20 response if the participant had ACR 20 observed for at least 2 consecutive study visits.
Time Frame: Day 169
Population: Analysis was carried out on the intent-to-treat (ITT) population defined as all randomized participants who received at least one dose of study medication. Two participants were unevaluable for response due to each missing 2 infusions of study drug.
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
participants | 129 | 26
Statistical Analysis 1: Comparison: Abatacept (ABA) vs Placebo (PLA); The first coprimary endpoint efficacy analysis tested for differences in ACR 20 response rate (RR) between the treatment arm receiving ABA plus background DMARDs and the treatment arm receiving placebo plus background DMARDs on Day 169. A 2-sided Cochran-Mantel-Haenszel (CMH) Chi-square test was used to compare these two treatment groups at the .05 level of significance, with stratification based on baseline history of anti-TNF status (current or prior use); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance was 5%. ACR 20 RR at 6 mos for PLA was expected to be ~25%. A sample of 256 in the ABA arm and 128 in PLA arm will yield a 96% power to detect a difference of 20% in ACR 20 at 5% significance level; All statistical tests and CI were 2-sided. Percentage of participants with response compared by estimate of weighted difference (Est of Weighted Diff); Est. Weighted. Diff: Day 169 ACR 20 = 30.8, 95% CI 2-sided [20.6 to 41.1] — Differences in ACR response between the two treatment groups represent the weighted average of the individual stratum differences

2. Primary Outcome: DB; Number of Participants Achieving Clinically Meaningful Improvement in Health Assessment Questionnaire (HAQ)
Description: The disability section of the full HAQ includes 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1= with some difficulty, 2= with much difficulty, and 3= unable to do. Higher scores= greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ response=an improvement of at least 0.3 units from baseline in HAQ disability Index.
Time Frame: Day 169
Population: Analysis was carried out on the intent-to-treat (ITT) population defined as all randomized subjects who received at least one dose of study medication. Two participants were unevaluable for response due to each missing 2 infusions of study drug.
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
participants | 121 | 31
Statistical Analysis 1: Comparison: Abatacept (ABA) vs Placebo (PLA); The two primary efficacy analyses tested first for differences in ACR 20 followed by testing HAQ response rates between the treatment arm receiving ABA plus background DMARDs and the treatment arm receiving PLA plus background DMARDs on Day 169. A 2-sided Cochran-Mantel-Haenszel (CMH) Chi-square test was used to compare these two treatment groups at the .05 level of significance, with stratification based on baseline history of anti-TNF status (current or prior use); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — If the ACR20 analysis was not significant (5% level), then the comparison for HAQ response was not undertaken. If ACR20 comparison was significant (5% level), then CMH Chi-square test compared HAQ response between groups (5% level); [statistical method as in outcome 1, analysis 1]; Est. of Weighted Diff: Day 169 HAQ = 24.0, 95% CI 2-sided [13.8 to 34.2] — All comparisons of changes from baseline and construction of confidence intervals for continuous measures were based on an ANCOVA model with treatment as the main factor and baseline value as covariate

3. Secondary Outcome: DB; Number of Participants With ACR 20, ACR 50, and ACR 70 Responses Over Time
Description: ACR 20/50/70 response requires a participant to have a 20/50/70% reduction in the number of swollen and tender joints, and a reduction of 20/50/70% in three of the following five parameters: physician global assessment of disease, participant global assessment of disease, participant assessment of pain, C-reactive protein or erythrocyte sedimentation rate, and degree of disability in Health Assessment Questionnaire (HAQ) score. A participant achieved a sustained ACR 20/50/70 response if the participant had ACR 20/50/70 observed for at least 2 consecutive study visits.
Time Frame: Days 15, 29, 57, 85, 113, 141, and 169
Population: Analysis was carried out on the intent-to-treat (ITT) population defined as all randomized subjects who received at least one dose of study medication. Two participants were unevaluable for response due to each missing 2 infusions of study drug. N=Number of Participants Analyzed, n=number of participants at visit
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
participants
  Day 15 ACR 20 | 45 | 7
  Day 15 ACR 50 | 6 | 0
  Day 15 ACR 70 | 2 | 0
  Day 29 ACR 20 | 84 | 25
  Day 29 ACR 50 | 22 | 4
  Day 29 ACR 70 | 6 | 1
  Day 57 ACR 20 | 118 | 32
  Day 57 ACR 50 | 34 | 9
  Day 57 ACR 70 | 13 | 0
  Day 85 ACR 20 | 118 | 24
  Day 85 ACR 50 | 46 | 8
  Day 85 ACR 70 | 15 | 1
  Day 113 ACR 20 | 126 | 31
  Day 113 ACR 50 | 46 | 5
  Day 113 ACR 70 | 20 | 0
  Day 141 ACR 20 | 141 | 26
  Day 141 ACR 50 | 65 | 6
  Day 141 ACR 70 | 26 | 0
  Day 169 ACR 20 | 129 | 26
  Day 169 ACR 50 | 52 | 5
  Day 169 ACR 70 | 26 | 2
Statistical Analysis 1: Comparison: Abatacept (ABA) vs Placebo (PLA); Differences in ACR 20 between the treatment arm receiving ABA plus background DMARDs and the treatment arm receiving PLA plus background DMARDs were compared using a 2-sided Cochran-Mantel-Haenszel (CMH) Chi-square test (.05 level of significance), with stratification based on baseline history of anti-TNF status (current or prior use); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; All statistical tests and CI were 2-sided. Percentage of participants with response compared by estimate of difference (Est of Diff); Est. of Diff: Day 15 ACR 20 = 12.3, 95% CI 2-sided [4.6 to 20.0]
Statistical Analysis 2: Comparison: Abatacept (ABA) vs Placebo (PLA); If ACR20 comparison was significant (5% level), then CMH Chi-square test compared ACR 50 response between groups (5% level). If the ACR20 analysis was not significant (5% level), then the comparison for ACR 50 response was not undertaken. A 2-sided Cochran-Mantel-Haenszel (CMH) Chi-square test was used to compare these two treatment groups at the .05 level of significance, with stratification based on baseline history of anti-TNF status (current or prior use); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 15 ACR 50 = 2.3, 95% CI 2-sided [-0.8 to 5.5]
Statistical Analysis 3: Comparison: Abatacept (ABA) vs Placebo (PLA); If ACR20 comparison was significant (5% level), then CMH Chi-square test compared ACR 70 response between groups (5% level). If the ACR20 analysis was not significant (5% level), then the comparison for ACR 70 response was not undertaken. A 2-sided Cochran-Mantel-Haenszel (CMH) Chi-square test was used to compare these two treatment groups at the .05 level of significance, with stratification based on baseline history of anti-TNF status (current or prior use); Test type: Superiority or Other; p = 0.784, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 15 ACR 70 = 0.8, 95% CI 2-sided [-1.3 to 2.9]
Statistical Analysis 4: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 29 ACR 20 = 14.0, 95% CI 2-sided [4.0 to 24.0]
Statistical Analysis 5: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.06, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 29 ACR 50 = 5.6, 95% CI 2-sided [-0.2 to 11.4]
Statistical Analysis 6: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.473, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 29 ACR 70 = 1.6, 95% CI 2-sided [-1.8 to 4.9]
Statistical Analysis 7: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 57 ACR 20 = 22.0, 95% CI 2-sided [11.3 to 32.8]
Statistical Analysis 8: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.076, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 57 ACR 50 = 6.5, 95% CI 2-sided [-0.6 to 13.7]
Statistical Analysis 9: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 57 ACR 70 = 5.1, 95% CI 2-sided [0.7 to 9.4]
Statistical Analysis 10: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 85 ACR 20 = 28.0, 95% CI 2-sided [17.4 to 38.7]
Statistical Analysis 11: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 85 ACR 50 = 12.0, 95% CI 2-sided [4.1 to 19.8]
Statistical Analysis 12: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.033, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 85 ACR 70 = 5.1, 95% CI 2-sided [0.4 to 9.8]
Statistical Analysis 13: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Est. of Diff: Day 113 ACR 20 = 25.9, 95% CI 2-sided [15.1 to 36.8]
Statistical Analysis 14: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Est. of Diff: Day 113 ACR 50 = 14.2, 95% CI 2-sided [6.6 to 21.9]
Statistical Analysis 15: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Est. of Diff: Day 113 ACR 70 = 7.8, 95% CI 2-sided [2.6 to 13.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 141 ACR 20 = 35.5, 95% CI 2-sided [24.6 to 46.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Est. of Diff: Day 141 ACR 50 = 20.9, 95% CI 2-sided [12.2 to 29.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Est. of Diff: Day 141 ACR 70 = 10.2, 95% CI 2-sided [4.4 to 16.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Est. of Diff: Day 169 ACR 20 = 30.8, 95% CI 2-sided [20.0 to 41.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Est. of Diff: Day 169 ACR 50 = 16.6, 95% CI 2-sided [8.6 to 24.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel; All statistical tests and CI were 2-sided. Percentage of participants with response compared by estimate of difference (Est of Weighted Diff); Est. of Diff: Day 169 ACR 70 = 8.7, 95% CI 2-sided [2.7 to 14.6] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: DB; Mean Time-matched Baseline Tender Joint Counts (TJCs) and Post-Baseline TJCs Over Time: ACR Core Component
Description: The mean TJC core component of the ACR scoring system was evaluated based on the number of tender joints in a standard 68 joint count, where an increasing number of tender joints indicates increasing level of severity. Time-matched baseline TJC values for each post-baseline TJC in the DB were presented for each visit and represent the mean baseline TJC value for only that cohort of participants with TJCs available at that visit.
Time Frame: BL
Population: Intent-to-treat (ITT) population: all randomized subjects receiving at least 1 dose of study drug. 2 participants were unevaluable for response due to each missing 2 infusions of study drug. N=total number of participants analyzed, n=the number of participants at time point with TJCs. Mean time-matched BL values reflect changing n-values over time.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
tender joints
  Day 15 cohort (n=251, n=126): baseline | 31.33 (12.86) | 32.75 (13.13)
  Day 15 cohort (n=251, n=126): post-baseline | 25.58 (14.39) | 30.35 (15.37)
  Day 29 cohort (n=248, n=128): baseline | 31.41 (13.11) | 32.72 (13.06)
  Day 29 cohort (n=248, n=128): post-baseline | 21.61 (14.53) | 27.52 (15.85)
  Day 57 cohort (n=251, n=129): baseline | 31.17 (12.90) | 32.31 (13.14)
  Day 57 cohort (n=251, n=129): post-baseline | 18.88 (14.41) | 24.20 (16.46)
  Day 85 cohort (n=249, n=129): baseline | 31.42 (13.05) | 32.58 (13.10)
  Day 85 cohort (n=249, n=129): post-baseline | 18.51 (14.15) | 25.56 (15.80)
  Day 113 cohort (n=246, n=128): baseline | 31.32 (13.10) | 32.65 (13.15)
  Day 113 cohort (n=246, n=128): post-baseline | 16.76 (14.18) | 25.21 (16.18)
  Day 141 cohort (n=252, n=128): baseline | 31.34 (13.10) | 32.28 (13.21)
  Day 141 cohort (n=252, n=128): post-baseline | 16.04 (13.89) | 23.67 (15.62)
  Day 169 cohort (n=254, n=130): baseline | 31.33 (13.06) | 32.43 (13.16)
  Day 169 cohort (n=254, n=130): post-baseline | 16.21 (13.94) | 25.55 (16.30)

5. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in TJC Over Time: ACR Core Component
Description: The mean TJC core component of the ACR scoring system was evaluated based on the number of tender joints in a standard 68 joint count, where an increasing number of tender joints indicates increasing level of severity. Mean Time-matched percentage of change from baseline = (time-matched baseline value - Post-baseline value)/time-matched baseline value x 100, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with TJCs available at that visit.
Time Frame: BL, Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=251, n=126) | 19.74 (2.19) | 6.43 (3.25)
  Day 29 cohort (n=248, n=128) | 32.68 (2.41) | 14.96 (3.84)
  Day 57 cohort (n=251, n=129) | 40.52 (2.56) | 24.99 (3.62)
  Day 85 cohort (n=249, n=129) | 40.40 (2.62) | 20.94 (3.49)
  Day 113 cohort (n=246, n=128) | 46.20 (2.76) | 21.72 (3.87)
  Day 141 cohort (n=252, n=128) | 49.06 (2.53) | 24.03 (4.05)
  Day 169 cohort (n=254, n=130) | 47.76 (2.66) | 20.04 (3.84)

6. Secondary Outcome: DB; Mean Time-matched Baseline Swollen Joint Count (SJC) and Post-Baseline SJCs Over Time: ACR Core Component
Description: The mean SJC core component of the ACR scoring system was evaluated based on the number of swollen joints in a standard 66 joint count, where an increasing number of swollen joints indicates increasing level of severity. Time-matched baseline SJC values for each post-baseline SJC in the DB were presented for each visit and represent the mean baseline SJC value for only that cohort of participants with SJCs available at that visit.
Time Frame: Days 15, 29, 57, 85, 113, 141, and 169
Population: Intent-to-treat (ITT) population: all randomized subjects receiving at least 1 dose of study drug. 2 participants were unevaluable for response due to each missing 2 infusions of study drug. N=total number of participants analyzed, n=the number of participants at time point with SJCs. Mean time-matched BL values reflect changing n-values over time.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
swollen joints
  Day 15 cohort (n=251, n=126): baseline | 22.31 (10.08) | 22.00 (9.79)
  Day 15 cohort (n=251, n=126): post-line | 17.88 (10.42) | 19.06 (10.97)
  Day 29 cohort (n=248, n=128): baseline | 22.49 (10.32) | 21.86 (9.79)
  Day 29 cohort (n=248, n=128): post-baseline | 15.55 (10.62) | 17.95 (11.83)
  Day 57 cohort (n=251, n=129): baseline | 22.15 (10.05) | 21.80 (9.78)
  Day 57 cohort (n=251, n=129): post-baseline | 13.44 (9.81) | 15.98 (10.17)
  Day 85 cohort (n=249, n=129): baseline | 22.42 (10.30) | 21.81 (9.77)
  Day 85 cohort (n=249, n=129): post-baseline | 12.44 (9.41) | 16.25 (11.92)
  Day 113 cohort (n=246, n=128): baseline | 22.48 (10.34) | 21.82 (9.81)
  Day 113 cohort (n=246, n=128): post-baseline | 12.18 (10.18) | 16.28 (10.78)
  Day 141 cohort (n=252, n=128): baseline | 22.38 (10.29) | 21.63 (9.74)
  Day 141 cohort (n=252, n=128): post-baseline | 11.06 (8.91) | 15.92 (10.49)
  Day 169 cohort (n=254, n=130): baseline | 22.35 (10.25) | 21.77 (9.75)
  Day 169 cohort (n=254, n=130): post-baseline | 12.00 (9.78) | 16.18 (11.10)

7. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in SJC Over Time: ACR Core Component
Description: The mean SJC core component of the ACR scoring system was evaluated based on the number of swollen joints in a standard 66 joint count, where an increasing number of swollen joints indicate increasing level of severity. Mean Time-matched percentage of change from baseline = (time-matched baseline value - Post-baseline value)/time-matched baseline value x 100, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with TJCs available at that visit.
Time Frame: Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=251, n=126) | 18.64 (2.38) | 13.13 (3.03)
  Day 29 cohort (n=248, n=128) | 32.68 (2.41) | 14.96 (3.84)
  Day 57 cohort (n=251, n=129) | 38.49 (2.70) | 24.98 (3.45)
  Day 85 cohort (n=249, n=129) | 44.42 (2.30) | 26.22 (3.72)
  Day 113 cohort (n=246, n=128) | 45.31 (2.75) | 22.87 (3.72)
  Day 141 cohort (n=252, n=128) | 49.38 (2.42) | 24.33 (3.77)
  Day 169 cohort (n=254, n=130) | 44.26 (2.84) | 23.78 (3.87)

8. Secondary Outcome: DB; Mean Time-matched Baseline Participant Pain Assessment Over Time: ACR Core Component
Description: The participant self-reported pain assessment is a core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale (VAS) with 0 mm representing no pain and 100 mm representing the most pain possible. For each post-baseline visit in the DB, time-matched baseline Participant Pain Assessment values were presented and represent the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: Intent-to-treat (ITT) population: all randomized subjects receiving at least 1 dose of study drug. 2 participants were unevaluable for response due to each missing 2 infusions of study drug. N=total number of participants analyzed, n=the number of participants at time point with data. Mean time-matched BL values reflect changing n-values over time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
units on a scale
  Day 15 cohort (n=247, n=126): baseline | 71.09 (19.57) | 69.20 (19.02)
  Day 15 cohort (n=247, n=126): post-baseline | 61.05 (22.45) | 67.65 (20.48)
  Day 29 cohort (n=240, n=128): baseline | 70.45 (19.77) | 69.80 (18.76)
  Day 29 cohort (n=240, n=128): post-baseline | 52.88 (23.93) | 61.07 (24.13)
  Day 57 cohort (n=246, n=129): baseline | 70.72 (19.70) | 69.26 (18.79)
  Day 57 cohort (n=246, n=129): post-baseline | 46.19 (25.26) | 55.91 (25.85)
  Day 85 cohort (n=245, n=129): baseline | 70.87 (19.85) | 69.40 (18.92)
  Day 85 cohort (n=245, n=129): post-baseline | 44.69 (26.13) | 60.16 (25.05)
  Day 113 cohort (n=239, n=126): baseline | 70.93 (19.71) | 70.27 (18.54)
  Day 113 cohort (n=239, n=126): post-baseline | 44.60 (26.19) | 60.17 (25.53)
  Day 141 cohort (n=249, n=127): baseline | 70.85 (19.73) | 69.34 (19.02)
  Day 141 cohort (n=249, n=127): post-baseline | 43.67 (27.20) | 59.80 (25.08)
  Day 169 cohort (n=251, n=130): baseline | 70.89 (19.67) | 69.47 (18.86)
  Day 169 cohort (n=251, n=130): post-baseline | 43.48 (27.76) | 62.21 (24.73)

9. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in Participant Pain Assessment Over Time: ACR Core Component
Description: Participant self-reported pain assessment is a core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale (VAS) with 0 mm representing no pain and 100 mm representing the most pain possible. Mean Time-matched percentage of change from baseline = (time-matched baseline value - Post-baseline value)/time-matched baseline value x 100, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL, Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 8
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=247, n=126) | 8.48 (3.82) | -3.19 (3.24)
  Day 29 cohort (n=240, n=128) | 18.31 (3.51) | 8.36 (3.26)
  Day 57 cohort (n=246, n=129) | 24.58 (6.39) | 16.65 (3.28)
  Day 85 cohort (n=245, n=129) | 26.76 (6.61) | 8.59 (3.79)
  Day 113 cohort (n=239, n=126) | 28.46 (4.79) | 9.87 (3.98)
  Day 141 cohort (n=249, n=127) | 27.29 (6.72) | 4.32 (5.55)
  Day 169 cohort (n=251, n=130) | 28.64 (5.70) | 4.36 (4.01)

10. Secondary Outcome: DB; Mean Time-matched Baseline HAQ-DI Over Time: ACR Core Component
Description: HAQ-DI is a self-administered questionnaire composed of 20 questions assessing physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. Questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The HAQ-DI is the weighted sum of the scale scores, with higher scores indicating poorer function. For each post-BL visit, time-matched BL HAQ-DI values were presented and represent the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
units on a scale
  Day 15 cohort (n=244, n=124): baseline | 1.84 (0.56) | 1.86 (0.56)
  Day 15 cohort (n=244, n=124): post-baseline | 1.69 (0.60) | 1.83 (0.56)
  Day 29 cohort (n=239, n=127): baseline | 1.84 (0.57) | 1.85 (0.56)
  Day 29 cohort (n=239, n=127): post-baseline | 1.59 (0.64) | 1.70 (0.62)
  Day 57 cohort (n=245, n=127): baseline | 1.83 (0.57) | 1.84 (0.55)
  Day 57 cohort (n=245, n=127): post-baseline | 1.49 (0.65) | 1.65 (0.63)
  Day 85 cohort (n=242, n=126): baseline | 1.84 (0.57) | 1.86 (0.56)
  Day 85 cohort (n=242, n=126): post-baseline | 1.45 (0.64) | 1.70 (0.63)
  Day 113 cohort (n=238, n=126): baseline | 1.85 (0.57) | 1.85 (0.56)
  Day 113 cohort (n=238, n=126): post-baseline | 1.44 (0.70) | 1.71 (0.64)
  Day 141 cohort (n=247, n=126): baseline | 1.84 (0.57) | 1.86 (0.56)
  Day 141 cohort (n=247, n=126): post-baseline | 1.41 (0.71) | 1.72 (0.64)
  Day 169 cohort (n=248, n=128): baseline | 1.84 (0.57) | 1.85 (0.56)
  Day 169 cohort (n=248, n=128): post-baseline | 1.38 (0.72) | 1.74 (0.63)

11. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in HAQ-DI Over Time: ACR Core Component
Description: A self-administered questionnaire with 20 questions assessing physical function in 8 domains:dressing,arising,eating,walking,hygiene,reach,grip and common activities.Questions evaluated on a 4-point scale:0=without any difficulty,1=with some difficulty,2=with much difficulty,and 3=unable to do. HAQ-DI=weighted sum of scale scores, with higher scores indicating poorer function. Mean time-matched % change from BL=(time-matched BL value - Post-BL value)/time-matched BL value x100, where time-matched BL value=the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 8
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=244, n=124) | 7.94 (1.45) | -1.10 (2.99)
  Day 29 cohort (n=239, n=127) | 13.75 (1.81) | 6.79 (2.49)
  Day 57 cohort (n=245, n=127) | 19.05 (1.78) | 9.61 (2.85)
  Day 85 cohort (n=242, n=126) | 21.00 (1.79) | 7.10 (2.68)
  Day 113 cohort (n=238, n=126) | 22.77 (1.98) | 5.96 (3.15)
  Day 141 cohort (n=247, n=126) | 24.41 (2.16) | 6.50 (2.68)
  Day 169 cohort (n=248, n=128) | 25.48 (2.14) | 5.08 (2.84)

12. Secondary Outcome: DB; Mean Time-matched Baseline Participant Global Assessment Over Time: ACR Core Component
Description: Participant self-reported global RA assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale (VAS) with 0 mm representing no pain and 100 mm representing the most pain possible. For each post-baseline visit in the DB, time-matched baseline Participant Global Assessment values were presented and represent the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
units on a scale
  Day 15 cohort (n=247, n=126): baseline | 69.30 (19.70) | 68.93 (20.38)
  Day 15 cohort (n=247, n=126): post-baseline | 58.55 (23.50) | 65.15 (21.38)
  Day 29 cohort (n=240, n=128): baseline | 68.86 (19.88) | 69.33 (20.03)
  Day 29 cohort (n=240, n=128): post-baseline | 52.48 (22.56) | 61.13 (24.42)
  Day 57 cohort (n=246, n=129): baseline | 69.02 (19.84) | 68.97 (20.10)
  Day 57 cohort (n=246, n=129): post-baseline | 45.07 (24.16) | 56.60 (26.03)
  Day 85 cohort (n=245, n=129): baseline | 69.40 (19.72) | 69.12 (20.23)
  Day 85 cohort (n=245, n=129): post-baseline | 43.27 (25.65) | 60.18 (24.88)
  Day 113 cohort (n=239, n=126): baseline | 69.40 (19.68) | 70.37 (19.15)
  Day 113 cohort (n=239, n=126): post-baseline | 45.05 (25.36) | 58.46 (25.61)
  Day 141 cohort (n=249, n=127): baseline | 69.09 (19.83) | 69.15 (20.36)
  Day 141 cohort (n=249, n=127): post-baseline | 43.72 (26.65) | 59.24 (25.69)
  Day 169 cohort (n=251, n=130): baseline | 69.22 (19.80) | 69.18 (20.16)
  Day 169 cohort (n=251, n=130): post-baseline | 43.51 (27.19) | 60.35 (25.69)

13. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in Participant Global Assessment Over Time: ACR Core Component
Description: Participant self-reported global RA assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100mm Visual Analog Scale (VAS) with 0mm representing no pain and 100mm representing the most pain possible. Mean Time-matched percentage of change from baseline = (time-matched baseline value - Post-baseline value)/time-matched baseline value x 100, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL, Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 8
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=247, n=126) | 11.54 (2.88) | -3.18 (4.48)
  Day 29 cohort (n=240, n=128) | 18.31 (2.93) | 2.13 (5.10)
  Day 57 cohort (n=246, n=129) | 29.84 (3.19) | 10.94 (4.70)
  Day 85 cohort (n=245, n=129) | 32.03 (4.08) | 2.89 (5.42)
  Day 113 cohort (n=239, n=126) | 30.83 (3.02) | 8.01 (5.48)
  Day 141cohort (n=249, n=127) | 29.46 (4.72) | 4.85 (5.51)
  Day 169 cohort (n=251, n=130) | 30.87 (4.10) | 4.52 (5.40)

14. Secondary Outcome: DB; Mean Time-matched Baseline Physician Global Assessment Over Time: ACR Core Component
Description: Physician global rheumatoid arthritis (RA) assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100mm Visual Analog Scale (VAS) with 0mm representing no pain and 100mm representing the most pain possible. For each post-baseline visit in the DB, time-matched baseline Physician Global Assessment values were presented and represent the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
units on a scale
  Day 15 cohort (n=250, n=126): baseline | 68.86 (17.40) | 66.91 (16.78)
  Day 15 cohort (n=250, n=126): post-baseline | 54.07 (21.93) | 61.43 (19.03)
  Day 29 cohort (n=246, n=126): baseline | 68.73 (17.41) | 66.81 (16.91)
  Day 29 cohort (n=246, n=126): post-baseline | 44.96 (21.03) | 53.71 (23.08)
  Day 57 cohort (n=252, n=127): baseline | 68.74 (17.34) | 66.92 (16.64)
  Day 57 cohort (n=252, n=127): post-baseline | 41.46 (21.93) | 49.21 (25.03)
  Day 85 cohort (n=247, n=124):baseline | 69.08 (17.42) | 66.81 (16.82)
  Day 85 cohort (n=247, n=124): post-baseline | 37.54 (21.29) | 53.06 (25.63)
  Day 113 cohort (n=246, n=127): baseline | 68.88 (17.26) | 67.45 (16.66)
  Day 113 cohort (n=246, n=127): post-baseline | 37.15 (21.88) | 54.49 (24.30)
  Day 141 cohort (n=252, n=127): baseline | 68.82 (17.39) | 67.03 (16.96)
  Day 141 cohort (n=252, n=127): post-baseline | 34.32 (21.56) | 51.58 (24.44)
  Day 169 cohort (n=254, n=129): baseline | 68.91 (17.40) | 67.05 (16.84)
  Day 169 cohort (n=254, n=129): post-baseline | 36.46 (23.65) | 52.37 (25.10)

15. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in Physician Global Assessment Over Time: ACR Core Component
Description: Physician global rheumatoid arthritis (RA) assessment core component of the ACR scoring system where increasing score indicates increasing level of severity as indicated on a 100mm Visual Analog Scale (VAS) with 0mm representing no pain and 100mm representing the most pain possible. Mean Time-matched percentage of change from baseline = (time-matched baseline value - Post-baseline value)/time-matched baseline value x 100, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL, Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 8
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=250, n=126) | 19.27 (2.45) | 6.26 (2.47)
  Day 29 cohort (n=246, n=126) | 32.32 (2.59) | 18.00 (3.08)
  Day 57 cohort (n=252, n=127) | 38.41 (2.38) | 25.51 (3.28)
  Day 85 cohort (n=247, n=124) | 43.74 (2.20) | 18.05 (4.04)
  Day 113cohort (n=246, n=127) | 45.11 (2.02) | 17.53 (3.26)
  Day 141 cohort (n=252, n=127) | 49.35 (1.89) | 21.34 (3.35)
  Day 169 cohort (n=254, n=129) | 45.18 (2.33) | 21.28 (3.14)

16. Secondary Outcome: DB; Mean Time-matched Baseline C-Reactive Protein (CRP) Levels Over Time: ACR Core Component
Description: CRP is an acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA) and a core component of the ACR scoring system. CRP was evaluated from serum samples. Increasing levels of CRP indicate increasing level of disease. For each post-baseline visit in the DB, time-matched baseline CRP values were presented and represent the mean baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
mg/dL
  Day 15 cohort (n=246, n=127): baseline | 4.53 (3.92) | 3.97 (3.57)
  Day 15 cohort (n=246, n=127): post-baseline | 3.20 (3.36) | 4.01 (3.54)
  Day 29 cohort (n=245, n=128): baseline | 4.62 (4.03) | 4.03 (3.62)
  Day 29 cohort (n=245, n=128): post-baseline | 2.70 (2.70) | 4.02 (3.63)
  Day 57 cohort (n=250, n=129): baseline | 4.60 (3.99) | 3.93 (3.58)
  Day 57 cohort (n=250, n=129): post-baseline | 2.39 (2.47) | 3.73 (4.06)
  Day 85 cohort (n=249, n=129): baseline | 4.59 (3.95) | 4.00 (3.61)
  Day 85 cohort (n=249, n=129): post-baseline | 2.36 (3.09) | 4.13 (4.11)
  Day 113 cohort (n=243, n=127): baseline | 4.62 (4.00) | 4.06 (3.62)
  Day 113 cohort (n=243, n=127): post-baseline | 2.26 (3.05) | 4.31 (4.62)
  Day 141 cohort (n=251, n=129): baseline | 4.62 (3.98) | 4.03 (3.60)
  Day 141 cohort (n=251, n=129): post-baseline | 2.20 (3.01) | 3.83 (4.17)
  Day 169 cohort (n=254, n=131): baseline | 4.60 (3.97) | 3.99 (3.59)
  Day 169 cohort (n=254, n=131): post-baseline | 2.31 (3.47) | 3.97 (4.19)

17. Secondary Outcome: DB; Mean Time-Matched Percentage of Change From Baseline in CRP Levels Over Time: ACR Core Component
Description: CRP is an acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA) and a core component of the ACR scoring system. CRP was evaluated from serum samples. Increasing levels indicate increasing level of disease. Mean Time-matched percentage of change from baseline = (time-matched baseline value - Post-baseline value)/time-matched baseline value x 100, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: Days 15, 29, 57, 85, 113, 141, and 169
Population: as for outcome 8
Measure: Mean (Standard Error); unit: percentage of change from BL
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
percentage of change from BL
  Day 15 cohort (n=246, n=127) | 14.03 (6.70) | -20.8 (8.24)
  Day 29 cohort (n=245, n=128) | 24.05 (4.20) | -20.1 (6.81)
  Day 57 cohort (n=250, n=129) | 22.83 (8.55) | -14.8 (8.23)
  Day 85 cohort (n=249, n=129) | 25.87 (9.68) | -31.9 (9.82)
  Day 113 cohort (n=243, n=127) | 34.52 (4.33) | -32.1 (10.37)
  Day 141 cohort (n=251, n=129) | 33.47 (4.76) | -22.8 (9.78)
  Day 169 cohort (n=254, n=131) | 25.05 (8.44) | -28.4 (11.82)

18. Secondary Outcome: DB; Mean Baseline Levels of Disease Biomarkers (Interleukin-6 (IL-6), Soluble IL-2 Receptor [sIL-2R], and Tumor Necrosing Factor [TNF]-Alpha) in Participants With Measurements at Day 169
Description: Potential biomarkers of disease (IL-6, SIL-2R, and TNF-Alpha) were determined from serum samples for all participants. The mean baseline value presented represents a time-matched Day 169 baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
pg/ml
  IL-6 (n=194, n=103) | 46.19 (62.49) | 43.18 (62.90)
  sIL-2R (n=193, n=88) | 1840 (767.0) | 1879 (1001)
  TNF-alpha (n=250, n=129) | 35.24 (73.17) | 30.64 (54.08)

19. Secondary Outcome: DB; Mean Change From Baseline to Day 169 in Levels of Disease Biomarkers (IL-6, sIL-2R, and TNF-alpha) in Participants With Measurements at Day 169
Description: The mean change from baseline in levels of potential biomarkers of disease (IL-6, SIL-2R, and TNF-Alpha) were determined from serum samples for all participants. Change from Baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with data available at Day 169.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
pg/ml
  IL-6 (n=194, n=103) | -24.4 (4.54) | 4.71 (8.13)
  sIL-2R (n=193, n=88) | -565 (40.40) | -36.1 (77.37)
  TNF-alpha (n=250, n=129) | -13.5 (4.06) | 5.87 (8.27)

20. Secondary Outcome: DB; Mean Baseline Levels of Disease Biomarkers (E-Selectin, Soluble Inter-Cellular Adhesion Molecule 1 [sICAM-1], and Matrix Metalloproteinase-3 [MMP-3]) in Participants With Measurements at Day 169
Description: Potential biomarkers of disease (E-selectin, sICAM-1, and MMP-3) were determined from serum samples for all participants. The mean baseline value presented represents a time-matched Day 169 baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
ng/ml
  E-selectin (n=190, n=103) | 93.03 (101.2) | 84.53 (71.64)
  sICAM-1 (n=187, n=103) | 426.6 (218.6) | 443.5 (327.1)
  MMP3 (n=192, n=133) | 86.53 (97.59) | 84.18 (133.5)

21. Secondary Outcome: DB; Mean Change From Baseline to Day 169 in Levels of Disease Biomarkers (E-Selectin, sICAM-1, and MMP-3) in Participants With Measurements at Day 169
Description: Potential biomarkers of disease (E-selectin, sICAM-1, and MMP-3) were determined from serum samples for all participants. Change from Baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with data available at Day 169.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
ng/ml
  E-selectin (n=190, n=103) | -10.6 (4.97) | 6.54 (4.34)
  sICAM-1 (n=187, n=103) | -22.2 (16.58) | -29.5 (20.17)
  MMP3 (n=192, n=133) | -37.0 (6.42) | -9.62 (11.51)

22. Secondary Outcome: DB; Mean Change From Baseline to Day 169 in Rheumatoid Factor (RF) Status
Description: Rheumatoid factor (RF or RhF) is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process. A positive value for RF was >20 IU/mL; a negative value for RF was ≤ 20 IU/mL.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
participants
  Baseline RF negative | 46 | 25
  Baseline RF negative change to RF positive | 3 | 3
  Baseline RF positive | 154 | 73
  Baseline RF positive change to RF negative | 13 | 0

23. Secondary Outcome: DB; Mean Baseline Short Form 36 (SF-36) Quality of Life Physical Component Summary (PCS), Mental Component Summary (MCS), and SF-36 Individual Component Scores For Participants With Measurements at Day 85
Description: SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Mean BL value presented represents a time-matched Day 85 BL value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
Units on a Scale
  PCS (n=243, n=128) | 27.41 (6.94) | 27.77 (6.31)
  MCS (n=243, n=128) | 41.13 (12.35) | 43.00 (11.94)
  Physical Function Scale Component (n=246, n=129) | 25.94 (8.90) | 26.31 (8.36)
  Role-Physical Scale Component (n=249, n=129) | 30.50 (6.25) | 31.96 (6.84)
  Bodily Pain Scale Component (n=248, n=129) | 30.49 (6.72) | 31.28 (6.64)
  General Health Scale Component (n=250, n=129) | 34.75 (9.18) | 34.95 (8.46)
  Vitality Scale Component (n=249, n=129) | 34.99 (8.51) | 36.70 (9.10)
  Social Functioning Scale Component (n=250, n=129) | 33.06 (10.78) | 33.95 (11.49)
  Role-Emotional Scale Component (n=249, n=128) | 35.79 (13.76) | 37.07 (13.83)
  Mental Health Scale Component (n=249, n=129) | 40.35 (12.75) | 42.72 (11.15)

24. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 85 in Short SF-36 PCS, MCS, and SF-36 Individual Component Scores
Description: SF-36 measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Change from Baseline= Post-baseline value - time-matched baseline value, where time-matched BL value = the mean BL value for only that cohort of participants with data available at Day 85.
Time Frame: BL, Day 85
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
Units on a Scale
  PCS (n=243, n=128) | 5.76 (0.52) | 2.12 (0.72)
  MCS (n=243, n=128) | 4.64 (0.63) | 2.08 (0.86)
  Physical Function Scale Component (n=246, n=129) | 3.97 (0.51) | 2.27 (0.71)
  Role-Physical Scale Component (n=249, n=129) | 5.88 (0.65) | 2.87 (0.90)
  Bodily Pain Scale Component (n=248, n=129) | 8.43 (0.55) | 2.81 (0.76)
  General Health Scale Component (n=250, n=129) | 3.65 (0.45) | 1.15 (0.62)
  Vitality Scale Component (n=249, n=129) | 5.49 (0.57) | 2.32 (0.80)
  Social Functioning Scale Component (n=250, n=129) | 6.83 (0.62) | 2.13 (0.87)
  Role-Emotional Scale Component (n=249, n=128) | 4.12 (0.83) | 3.14 (1.16)
  Mental Health Scale Component (n=249, n=129) | 4.29 (0.58) | 1.70 (0.80)
Statistical Analysis 1: Comparison: Abatacept (ABA) vs Placebo (PLA); Differences in mean changes from baseline between the 2 treatment groups (ABA and PLA) in PCS, MCS, and the 8 subscale scores at Day 85 were compared using ANCOVA models. Adjusted difference (Adj Diff) from PLA group with 95% CIs and p-values were calculated, and adjustment was based on ANCOVA model with treatment group as factor and baseline value as covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 85 PCS = 3.63, 95% CI 2-sided [1.89 to 5.38]
Statistical Analysis 2: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA; Adj Diff: Day 85 MCS = 2.57, 95% CI 2-sided [0.47 to 4.67]
Statistical Analysis 3: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.052, ANCOVA; Adj Diff: Day 85 Physical Function = 1.70, 95% CI 2-sided [-0.01 to 3.41]
Statistical Analysis 4: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA; Adj Diff: Day 85 Role-Physical = 3.01, 95% CI 2-sided [0.83 to 5.19]
Statistical Analysis 5: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 85 Bodily Pain = 5.62, 95% CI 2-sided [3.77 to 7.47]
Statistical Analysis 6: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA; Adj Diff: General Health = 2.51, 95% CI 2-sided [0.99 to 4.02]
Statistical Analysis 7: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA; Adj Diff: Day 85 Vitality = 3.17, 95% CI 2-sided [1.24 to 5.10]
Statistical Analysis 8: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 85 Social Functioning = 4.69, 95% CI 2-sided [2.59 to 6.79]
Statistical Analysis 9: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.494, ANCOVA; Adj Diff: Day 85 Role Emotional = 0.97, 95% CI 2-sided [-1.82 to 3.77]
Statistical Analysis 10: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA; Adj Diff: Day 85 Mental Health = 2.59, 95% CI 2-sided [0.65 to 4.54]

25. Secondary Outcome: DB; Mean Baseline SF-36 PCS, MCS, and SF-36 Individual Component Scores For Participants With Measurements at Day 169
Description: SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Mean BL value presented represents a time-matched Day 169 BL value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
Units on a Scale
  PCS (n=242, n=129) | 27.36 (6.88) | 27.75 (6.29)
  MCS (n=242, n=129) | 41.56 (12.33) | 42.98 (11.90)
  Physical Function Scale Component (n=247, n=130) | 25.96 (8.88) | 26.24 (8.37)
  Role-Physical Scale Component (n=249, n=130) | 30.56 (6.29) | 31.93 (6.82)
  Bodily Pain Scale Component (n=248, n=130) | 30.54 (6.76) | 31.27 (6.62)
  General Health Scale Component (n=252, n=130) | 34.81 (9.20) | 35.05 (8.51)
  Vitality Scale Component (n=252, n=130) | 35.07 (8.52) | 36.69 (9.06)
  Social Functioning Scale Component (n=251, n=130) | 33.17 (10.81) | 33.84 (11.52)
  Role-Emotional Scale Component (n=249, n=129) | 35.96 (13.77) | 36.97 (13.83)
  Mental Health Scale Component (n=252, n=130) | 40.50 (12.81) | 42.80 (11.14)

26. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 169 in SF-36 PCS, MCS, and SF-36 Individual Component Scores For Participants With Measurements at Day 169
Description: SF-36 measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Change from Baseline= Post-baseline value - time-matched baseline value, where time-matched BL value = the mean BL value for only that cohort of participants with data available at Day 169.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
Units on a Scale
  PCS (n=242, n=129) | 6.58 (0.55) | 1.12 (0.75)
  MCS (n=242, n=129) | 5.15 (0.64) | 2.11 (0.87)
  Physical Function Scale Component (n=247, n=130) | 5.30 (0.58) | 1.27 (0.80)
  Role-Physical Scale Component (n=249, n=130) | 6.52 (0.63) | 1.29 (0.87)
  Bodily Pain Scale Component (n=248, n=130) | 8.72 (0.56) | 2.48 (0.77)
  General Health Scale Component (n=252, n=130) | 4.02 (0.48) | 0.74 (0.67)
  Vitality Scale Component (n=252, n=130) | 6.55 (0.60) | 1.77 (0.83)
  Social Functioning Scale Component (n=251, n=130) | 7.31 (0.65) | 2.39 (0.91)
  Role-Emotional Scale Component (n=249, n=129) | 6.00 (0.83) | 2.46 (1.15)
  Mental Health Scale Component (n=252, n=130) | 4.31 (0.56) | 1.61 (0.79)
Statistical Analysis 1: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 PCS = 5.46, 95% CI 2-sided [3.64 to 7.29]
Statistical Analysis 2: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA; Adj Diff: Day 169 MCS = 3.04, 95% CI 2-sided [0.91 to 5.17]
Statistical Analysis 3: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 Physical Function = 4.03, 95% CI 2-sided [2.08 to 5.98]
Statistical Analysis 4: Comparison: Placebo (PLA); Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 Role-Physical = 5.22, 95% CI 2-sided [3.10 to 7.35]
Statistical Analysis 5: Comparison: Abatacept (ABA) vs Placebo (PLA); Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 Bodily Pain = 6.24, 95% CI 2-sided [4.37 to 8.11]
Statistical Analysis 6: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 General Health = 3.27, 95% CI 2-sided [1.64 to 4.90]
Statistical Analysis 7: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 Vitality = 4.78, 95% CI 2-sided [2.76 to 6.79]
Statistical Analysis 8: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj Diff: Day 169 Social Functioning = 4.92, 95% CI 2-sided [2.71 to 7.12]
Statistical Analysis 9: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.013, ANCOVA; Adj Diff: Day 169 Role Emotional = 3.54, 95% CI 2-sided [0.74 to 6.33]
Statistical Analysis 10: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.006, ANCOVA; Adj Diff: Mental Health = 2.70, 95% CI 2-sided [0.79 to 4.60]

27. Secondary Outcome: DB; Mean Baseline HAQ-DI and HAQ Component Scores in Participants With Assessments at Day 169
Description: The HAQ DI is a self-administered questionnaire composed of 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. Questions are evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. HAQ-DI is a weighted sum of the scale scores, with a higher score indicating poorer function. The mean baseline value presented represents a time-matched Day 169 baseline value for only that cohort of participants with assessments available at that visit.
Time Frame: BL
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
units on a scale
  HAQ-DI (n=249, n=130) | 1.83 (0.58) | 1.82 (0.60)
  HAQ dressing and grooming (n=214, n=97) | 1.64 (0.75) | 1.54 (0.69)
  HAQ arising (n=214, n=97) | 1.42 (0.72) | 1.43 (0.73)
  HAQ eating (n=214, n=97) | 1.76 (0.83) | 1.78 (0.87)
  HAQ walking (n=213, n=95) | 1.56 (0.70) | 1.51 (0.76)
  HAQ hygiene (n=213, n=97) | 2.14 (0.88) | 2.21 (0.87)
  HAQ reaching (n=213, n=97) | 2.04 (0.79) | 1.97 (0.87)
  HAQ gripping (n=212, n=97) | 1.96 (0.53) | 1.93 (0.62)
  HAQ activities (n=213, n=97) | 2.00 (0.79) | 1.95 (0.86)

28. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 169 in HAQ-DI and HAQ Component Scores in Participants With Assessments at Day 169
Description: HAQ DI is a self-administered questionnaire composed of 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. Questions evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. HAQ-DI=weighted sum of the scale scores. Higher score indicates poorer function.Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at Day 169.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
units on a scale
  HAQ-DI (n=249, n=130) | -0.45 (0.03) | -0.11 (0.04)
  HAQ dressing and grooming (n=214, n=97) | -0.58 (0.05) | -0.26 (0.07)
  HAQ arising (n=214, n=97) | -0.61 (0.04) | -0.29 (0.07)
  HAQ eating (n=214, n=97) | -0.54 (0.05) | -0.07 (0.07)
  HAQ walking (n=213, n=95) | -0.50 (0.05) | -0.24 (0.07)
  HAQ hygiene (n=213, n=97) | -0.28 (0.05) | -0.05 (0.07)
  HAQ reaching (n=213, n=97) | -0.54 (0.05) | -0.11 (0.08)
  HAQ gripping (n=212, n=97) | -0.47 (0.05) | -0.15 (0.07)
  HAQ activities (n=213, n=97) | -0.48 (0.05) | -0.08 (0.07)
Statistical Analysis 1: Comparison: Abatacept (ABA) vs Placebo (PLA); Mean changes from baseline in HAQ disability index were compared between treatment groups using analysis of covariance (ANCOVA) models and 95% confidence intervals were calculated. This analysis was based on the LOCF data set. Similar analyses were also conducted for each of the 8 individual categories: 1) dressing and grooming; 2) arising; 3) eating; 4) walking; 5) hygiene; 6) reach; 7) grip; and 8) common daily activities. Adjusted Mean Change From Baseline = Adj M Chg From BL; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: HAQ-DI = -0.34, 95% CI 2-sided [-0.44 to -0.23]
Statistical Analysis 2: Comparison: Abatacept (ABA) vs Placebo (PLA); Mean changes from baseline in HAQ disability index were compared between treatment groups using analysis of covariance (ANCOVA) models and 95% confidence intervals were calculated. This analysis was based on the LOCF data set. Similar analyses were also conducted for each of the 8 individual categories: 1) dressing and grooming; 2) arising; 3) eating; 4) walking; 5) hygiene; 6) reach; 7) grip; and 8) common daily activities. Adjusted Mean Change From Baseline= Adj M Chg From BL; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: Dressing and Grooming = -0.32, 95% CI 2-sided [-0.49 to -0.14]
Statistical Analysis 3: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: Arising = -0.32, 95% CI 2-sided [-0.47 to -0.16]
Statistical Analysis 4: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: Eating = -0.48, 95% CI 2-sided [-0.65 to -0.30]
Statistical Analysis 5: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA; Adj M Chg from BL: Walking = -0.26, 95% CI 2-sided [-0.44 to -0.09]
Statistical Analysis 6: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 2]; Test type: Superiority or Other; p = 0.010, ANCOVA; Adj M Chg from BL: Hygiene = -0.22, 95% CI 2-sided [-0.39 to -0.05]
Statistical Analysis 7: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: Reaching = -0.43, 95% CI 2-sided [-0.61 to -0.25]
Statistical Analysis 8: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: Gripping = -0.32, 95% CI 2-sided [-0.49 to -0.15]
Statistical Analysis 9: Comparison: Abatacept (ABA) vs Placebo (PLA); [analysis description as in outcome 28, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; Adj M Chg from BL: Activities = -0.40, 95% CI 2-sided [-0.58 to -0.22]

29. Secondary Outcome: DB; Mean Disease Activity Score (DAS)28 (C-Reactive Protein [CRP]) and Mean Disease Activity Score (Erythrocyte Sedimentation Rate [ESR]) at Day 169
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP levels, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline. The mean BL value presented represents a time-matched Day 169 BL value for only that cohort of participants with assessments available at that visit.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
Units on a Scale
  Baseline DAS28 (CRP); n=251, n=130 | 6.53 (0.89) | 6.51 (0.78)
  Day 169 DAS28 (CRP); n=251, n=130 | 4.70 (1.45) | 5.78 (1.33)
  Baseline DAS28 (ESR); n=182, n=98 | 6.88 (0.99) | 6.88 (0.92)
  Day 169 DAS28 (ESR); n=182, n=98 | 4.90 (1.55) | 6.17 (1.34)

30. Secondary Outcome: DB; Adjusted Mean Change From Baseline to Day 169 in DAS28 (CRP) and DAS28 (ESR)
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at Day 169.
Time Frame: BL, Day 169
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 133
Units on a Scale
  DAS28 (CRP); n=251, n=130 | -1.83 (0.08) | -0.74 (0.11)
  DAS28 (ESR); n=182, n=98 | -1.98 (0.10) | -0.71 (0.14)

31. Secondary Outcome: DB; Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, or AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.Related AE/SAE=Certain,Probable,Possible,or Missing relationship to Drug
Time Frame: From BL up to database lock for DB period (6/2/2004)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 258 | 133
participants
  Deaths | 1 | 0
  SAEs | 27 | 15
  Related SAEs | 7 | 1
  SAEs Leading to Discontinuation | 7 | 2
  AEs | 205 | 95
  Related AEs | 107 | 39
  AEs Leading to Discontinuation | 9 | 4

32. Secondary Outcome: DB; Number of Participants AEs of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections, serious infections, and opportunistic infections; autoimmune disorders; neoplasms; acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion) and peri-infusional AEs (pre-specified AEs occurring within 24 hours of the start of infusion).
Time Frame: From BL up to database lock for DB period (6/2/2004)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 258 | 133
participants
  Infections | 97 | 43
  Neoplasms | 7 | 1
  Pre-specified autoimmune disorders | 4 | 0
  Acute infusional AEs | 13 | 4
  Peri-infusional AEs | 40 | 17

33. Secondary Outcome: DB; Number of Participants With Hematology Laboratories Meeting Marked Abnormality (MA) Criteria
Description: Upper Normal Limit (ULN), Lower Normal Limit (LLN), Baseline (BL). Marked abnormality criteria are: Hemoglobin (HGB): >3 g/dL decrease from BL; Hematocrit: <0.75 * BL; Erythrocytes: <0.75 * BL; Platelets (PLT): <0.67 * LLN/>1.5 * ULN, or if BL < LLN then use 0.5 * BL/<100,000 mm^3; Leukocytes: <0.75 * LLN/ >1.25 * ULN, or if BL<LLN then use <0.8 * BL/>ULN, or if BL>ULN then use >1.2 * BL/<LLN; neutrophils+bands: <1.0 * 10^3 c/uL; eosinophils: >0.750 * 10^3 c/uL; basophils: > 400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750 * 10^3 c/uL/ >7.50 * 10^3 c/uL.
Time Frame: From BL up to database lock for DB period (6/2/2004)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 131
participants
  Low HGB (LLN=11.5 g/dL) | 0 | 1
  Low hematocrit (LLN=34%) | 0 | 1
  Low erythrocytes (LLN=3.8 x10*6 cells/μL) | 0 | 0
  Low PLT (LLN=140*10^9 cells/μL) | 1 | 1
  High PLT (ULN=450*10^9 cells/L) | 1 | 0
  Low leukocytes (LLN= 3.8*10^3 cells/μL) | 2 | 0
  High leukocytes (ULN = 10.6*10^3 cells/μL) | 18 | 14
  Low neutrophils+bands(LLN=1.8*10^3 cells/μL) | 0 | 0
  Low lymphocytes (LLN= 0.7*10^3 cells/μL) | 0 | 0
  High lymphocytes(ULN=4.5*10^3 cells/μL) | 0 | 0
  High monocytes (ULN=1*10^3 cells/μL) | 0 | 0
  High basophils (ULN= 0.2*10^3 cells/μL) | 0 | 0
  High eosinophils (ULN= 7*10^3 cells/μL) | 0 | 0

34. Secondary Outcome: DB; Number of Participants With Blood Chemistry Laboratories Meeting MA Criteria
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2* ULN, or if BL>ULN then use >3* BL; aspartate aminotransferase (AST): >3* ULN, or if BL>ULN then use >4* BL; alanine aminotransferase (ALT): >3* ULN, or if BL>ULN then use >4* BL; G-Glutamyl transferase (GGT): >2* ULN, or if BL>ULN then use >3* BL; Bilirubin: >2* ULN, or if BL>ULN then use >4* BL; blood urea nitrogen (BUN): >2* BL; creatinine: >1.5* BL
Time Frame: From BL up to database lock for DB period (6/2/2004)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Abatacept (ABA) | Placebo (PLA)
Number analyzed (Participants) | 256 | 131
participants
  High ALP (ULN=400 U/L) | 0 | 0
  High AST (ULN=44 U/L) | 2 | 2
  High ALT (ULN=55 U/L) | 4 | 1
  High GGT (ULN=65 U/L) | 0 | 0
  High bilirubin (ULN=1.2 mg/dL) | 0 | 0
  High BUN (ULN=26 mg/dL) | 0 | 0
  High creatinine (ULN=1.5 mg/dL) | 11 | 5

35. Primary Outcome: Open-Label Period (OL); Number of Participants With Death, Serious Adverse Events (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs, Related AEs, or AEs Leading to Discontinuation
Description: as for outcome 31
Time Frame: From first day of OL to 5.5 years
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Open-label ABA
Number analyzed (Participants) | 317
participants
  Deaths | 6
  SAEs | 136
  Related SAEs | 24
  SAEs Leading to Discontinuation | 20
  AEs | 302
  Related AEs | 192
  AEs Leading to Discontinuation | 34

36. Secondary Outcome: DB; Number of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Responses by Enzyme-Linked Immunosorbant Assay (ELISA)
Description: Serum samples from all treated adult participants with active rheumatoid arthritis (RA) were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: From BL to Day 169
Population: All treated participants in the double-blind period with at least 1 post-baseline immunogenicity result
Measure: Number; unit: participants
Groups:
- All Treated DB Participants: Participants with active RA who met the inclusion/exclusion criteria for this study were randomized to receive either abatacept or placebo on a background of DMARDs. Participants must have been treated with anti-TNF therapy for at least 3 months and designated as anti-TNF therapy failures due to inadequate efficacy. Participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of abatacept. Abatacept or placebo was administered on Days 1, 15, 29 and every 28 days thereafter for a total of 7 doses. Each dose was infused intravenously over approximately 30 minutes.
Arm/Group | All Treated DB Participants
Number analyzed (Participants) | 234
participants
  Anti-abatacept antibodies | 1
  Anti-CTLA4 antibodies | 2
  Total | 3

37. Primary Outcome: OL; Number of Participants AEs of Special Interest
Description: as for outcome 32
Time Frame: From first day of OL to 5.5 years
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Open-label ABA
Number analyzed (Participants) | 317
participants
  Infections | 254
  Neoplasms (benign, malignant, and unspecified) | 42
  Malignancies | 21
  Pre-specified autoimmune disorders | 17
  Acute infusional AEs | 65
  Peri-infusional AEs | 22

38. Primary Outcome: OL; Number of Participants With Hematology Laboratories Meeting Marked Abnormality Criteria
Description: as for outcome 33
Time Frame: From first day of OL to 5.5 years
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Open-label ABA
Number analyzed (Participants) | 315
participants
  Low HGB (LLN=11.5 g/dL) | 12
  Low hematocrit (LLN=34%) | 18
  Low erythrocytes (LLN=3.8 x10*6 cells/μL) | 9
  Low PLT (LLN=140*10^9 cells/L) | 8
  High PLT (ULN=450*10^9 cells/L) | 1
  Low leukocytes (LLN=3.8*10^3 cells/μL) | 6
  High leukocytes (ULN=10.6*10^3 c/μL) | 49
  Low neutrophils + bands (LLN=1.8*10^3 c/μL)) | 2
  Low lymphocytes (LLN=0.7*10^3 cells/μL) | 61
  High lymphocytes (ULN=4.5*10^3 cells/μL) | 0
  High monocytes (ULN=1*10^3 cells/μL) | 2
  High basophils (ULN=0.2*10^3 cells/μL) | 0
  High eosinophils (ULN=7*10^3 cells/μL) | 31

39. Primary Outcome: OL; Number of Participants With Blood Chemistry Laboratories Meeting Marked Abnormality Criteria
Description: as for outcome 34
Time Frame: From first day of OL to 5.5 years
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Open-label ABA
Number analyzed (Participants) | 315
participants
  High ALP (ULN=400 U/L) | 3
  High AST (ULN=44 U/L) | 12
  High ALT (ULN=55 U/L) | 12
  High GGT (ULN=65 U/L) | 30
  High bilirubin (ULN=1.2 mg/dL) | 2
  High BUN (ULN=26 mg/dL) | 20
  High creatinine (ULN=1.5 mg/dL) | 77

40. Primary Outcome: OL; Mean Time-matched Baseline Immunoglobulin (Ig) Levels Over the OL
Description: Serum samples collected from participants were used to determine serum levels of IgA, IgM, and IgG. Time-matched baseline values were presented by visit and represented the mean baseline value for only that cohort of participants with serum samples available at that visit.
Time Frame: Baseline and Days 169, 365, 729, and 1093
Population: All treated participants with available serum samples. N=the total number of participants analyzed, n=the number of participants at that time point with available serum samples. Mean time-matched baseline values reflect changing n-values over time.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- OL: ABA: Participants treated in the OL who were randomized to receive placebo on a background of DMARDs in the DB. Participants weighing > 100 kg received 1 g, participants weighing ≥ 60 kg and ≤ 100 kg received 750 mg, and participants weighing < 60 kg received 500 mg on a background of DMARDs IV on Days 1, 15, 29, 57, 85, 113, and 141.
- OL: PLA: Participants treated in the OL who were randomized to receive placebo on a background of DMARDs in the DB. Placebo was administered IV on Days 1, 15, 29, 57, 85, 113, and 141.
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 201 | 96
mg/dL
  Day 169 cohort (n=201, n=96): IgA | 327.9 (170.8) | 326.9 (203.3)
  Day 169 cohort (n=201, n=96): IgG | 1346.0 (473.0) | 1364.0 (532.2)
  Day 169 cohort (n=201, n=96): IgM | 180.1 (128.3) | 160.1 (86.91)
  Day 365 cohort (n=182, n=84): IgA | 337.6 (173.0) | 318.6 (204.4)
  Day 365 cohort (n=182, n=84): IgG | 1320.0 (421.2) | 1341.0 (525.9)
  Day 365 cohort (n=182, n=84): IgM | 175.7 (113.5) | 159.5 (88.33)
  Day 729 cohort (n=163, n=75): IgA | 322.2 (156.8) | 327.6 (218.5)
  Day 729 cohort (n=163, n=75): IgG | 1337.0 (421.4) | 1338.0 (528.7)
  Day 729 cohort (n=163, n=75): IgM | 184.1 (137.0) | 165.9 (91.12)
  Day 1093 cohort (n=76, n=42): IgG | 294.1 (128.6) | 329.6 (167.8)
  Day 1093 cohort (n=76, n=42): IgG | 1374.0 (537.3) | 1478.0 (562.9)
  Day 1093 cohort (n=76, n=42): IgM | 175.5 (158.1) | 174.2 (89.43)

41. Primary Outcome: OL; Mean Time-matched Change From Baseline in Immunoglobulin (Ig) Levels Over the OL
Description: Serum samples collected from participants were used to determine serum levels of IgA, IgM, and IgG. Time-matched mean change from baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with serum samples available at that visit.
Time Frame: BL, Days 169, 365, 729, and 1093
Population: as for outcome 40
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 201 | 96
mg/dL
  Day 169 cohort (n=201, n=96): IgA | -35.3 (3.61) | 1.10 (8.12)
  Day 169 cohort (n=201, n=96): IgG | -233.0 (19.54) | -72.8 (35.74)
  Day 169 cohort (n=201, n=96): IgM | -17.8 (3.59) | -5.42 (3.63)
  Day 365 cohort (n=182, n=84): IgA | -37.5 (4.93) | -33.0 (10.12)
  Day 365 cohort (n=182, n=84): IgG | -282.0 (18.60) | -251.0 (39.41)
  Day 365 cohort (n=182, n=84): IgM | -23.0 (4.21) | -18.3 (4.21)
  Day 729 cohort (n=163, n=75): IgA | -37.3 (6.13) | -30.0 (10.42)
  Day 729 cohort (n=163, n=75): IgG | -344.0 (2.81) | -257.0 (38.30)
  Day 729 cohort (n=163, n=75): IgM | -19.4 (6.01) | -16.1 (6.02)
  Day 1093 cohort (n=76, n=41): IgA | -35.6 (7.50) | -69.4 (16.83)
  Day 1093 cohort (n=76, n=42): IgG | -396.0 (46.77) | -377.0 (55.94)
  Day 1093 cohort (n=76, n=42): IgM | -29.7 (9.03) | -24.7 (9.51)

42. Secondary Outcome: OL; Number of Participants With ACR 20, ACR 50, and ACR 70 Responses Over Time For Participants Treated in the OL
Description: as for outcome 3
Time Frame: Days 15, 29, 57, 85, 113, 141, 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1261, 1457, 1625, and 1821
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 214 | 98
participants
  Day 15 ACR 20 (n=214, n=97) | 43 | 6
  Day 15 ACR 50 (n=213, n=97) | 5 | 0
  Day 15 ACR 70 (n=214, n=97) | 1 | 0
  Day 29 ACR 20 (n=210, n=97) | 77 | 23
  Day 29 ACR 50 (n=213, n=97) | 20 | 4
  Day 29 ACR 70 (n=213, n=97) | 4 | 1
  Day 57 ACR 20 (n=211, n=98) | 109 | 30
  Day 57 ACR 50 (n=213, n=98) | 31 | 9
  Day 57 ACR 70 (n=213, n=98) | 11 | 0
  Day 85 ACR 20 (n=211, n=97) | 113 | 22
  Day 85 ACR 50 (n=211, n=97) | 44 | 8
  Day 85 ACR 70 (n=212, n=98) | 15 | 1
  Day 113 ACR 20 (n=203, n=95) | 120 | 31
  Day 113 ACR 50 (n=206, n=97) | 42 | 5
  Day 113 ACR 70 (n=206, n=97) | 20 | 0
  Day 141 ACR 20 (n=212, n=96) | 136 | 26
  Day 141 ACR 50 (n=214, n=97) | 62 | 6
  Day 141 ACR 70 (n=214, n=97) | 25 | 0
  Day 169 ACR 20 (n=208, n=98) | 125 | 26
  Day 169 ACR 50 (n=209, n=98) | 50 | 5
  Day 169 ACR 70 (n=212, n=98) | 25 | 2
  Day 253 ACR 20 (n=203, n=95) | 127 | 49
  Day 253 ACR 50 (n=199, n=97) | 58 | 28
  Day 253 ACR 70 (n=204, n=98) | 25 | 10
  Day 365 ACR 20 (n=198, n=96) | 129 | 63
  Day 365 ACR 50 (n=201, n=95) | 65 | 37
  Day 365 ACR 70 (n=202, n=96) | 37 | 13
  Day 449 ACR 20 (n=181, n=82) | 124 | 61
  Day 449 ACR 50 (n=181, n=85) | 73 | 37
  Day 449 ACR 70 (n=182, n=85) | 32 | 18
  Day 533 ACR 20 (n=168, n=76) | 115 | 53
  Day 533 ACR 50 (n=169, n=77) | 71 | 30
  Day 533 ACR 70 (n=171, n=78) | 36 | 10
  Day 617 ACR 20 (n=163, n=72) | 120 | 55
  Day 617 ACR 50 (n=161, n=70) | 73 | 32
  Day 617 ACR 70 (n=162, n=71) | 33 | 13
  Day 729 ACR 20 (n=156, n=71) | 117 | 49
  Day 729 ACR 50 (n=153, n=72) | 70 | 30
  Day 729 ACR 70 (n=155, n=74) | 35 | 13
  Day 813 ACR 20 (n=140, n=60) | 105 | 47
  Day 813 ACR 50 (n=141, n=61) | 62 | 23
  Day 813 ACR 70 (n=143, n=62) | 28 | 6
  Day 897 ACR 20 (n=134, n=62) | 107 | 45
  Day 897 ACR 50 (n=137, n=61) | 64 | 29
  Day 897 ACR 70 (n=138, n=62) | 27 | 8
  Day 981 ACR 20 (n=140, n=57) | 104 | 40
  Day 981 ACR 50 (n=143, n=58) | 66 | 25
  Day 981 ACR 70 (n=140, n=60) | 31 | 9
  Day 1093 ACR 20 (n=134, n=55) | 109 | 44
  Day 1093 ACR 50 (n=137, n=57) | 70 | 29
  Day 1093 ACR 70 (n=137, n=58) | 32 | 16
  Day 1261 ACR 20 (n=126, n=52) | 99 | 42
  Day 1261 ACR 50 (n=126, n=53) | 60 | 24
  Day 1261 ACR 70 (n=130, n=55) | 27 | 15
  Day 1457 ACR 20 (n=115, n=50) | 87 | 41
  Day 1457 ACR 50 (n=115, n=50) | 53 | 24
  Day 1457 ACR 70 (n=118, n=50) | 22 | 11
  Day 1625 ACR 20 (n=110, n=49) | 89 | 33
  Day 1625 ACR 50 (n=111, n=48) | 50 | 19
  Day 1625 ACR 70 (n=112, n=49) | 26 | 12
  Day 1821 ACR 20 (n=106, n=46) | 81 | 35
  Day 1821 ACR 50 (n=106, n=47) | 55 | 24
  Day 1821 ACR 70 (n=109, n=47) | 24 | 10

43. Secondary Outcome: OL; Number of Participants With Low Disease Activity (LDAS) or Remission For Participants Treated in the OL
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). A clinically significant response= decrease in DAS28 score of >1.2 from baseline.
Time Frame: Days 15, 29, 57, 85, 113, 141, 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1261, 1457, 1625, and 1821
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 213 | 98
participants
  Day 15 LDAS (n=209, n=95) | 5 | 0
  Day 15 Remission (n=209, n=95) | 1 | 0
  Day 29 LDAS (n=206, n=96) | 10 | 1
  Day 29 Remission (n=206, n=96) | 5 | 1
  Day 57 LDAS (n=210, n=97) | 19 | 5
  Day 57 Remission (n=210, n=97) | 11 | 1
  Day 85 LDAS (n=212, n=98) | 22 | 4
  Day 85 Remission (n=212, n=98) | 11 | 3
  Day 113 LDAS (n=202, n=93) | 28 | 4
  Day 113 Remission (n=202, n=93) | 11 | 0
  Day 141 LDAS (n=213, n=96) | 41 | 4
  Day 141 Remission (n=213, n=96) | 15 | 2
  Day 169 LDAS (n=208, n=96) | 38 | 5
  Day 169 Remission (n=208, n=96) | 23 | 1
  Day 253 LDAS (n=195, n=89) | 33 | 19
  Day 253 Remission (n=195, n=89) | 19 | 12
  Day 365 LDAS (n=194, n=93) | 47 | 22
  Day 365 Remission (n=194, n=93) | 27 | 17
  Day 449 LDAS (n=170, n=76) | 48 | 25
  Day 449 Remission (n=170, n=76) | 24 | 15
  Day 533 LDAS (n=164, n=73) | 46 | 21
  Day 533 Remission (n=164, n=73) | 26 | 13
  Day 617 LDAS (n=164, n=69) | 51 | 23
  Day 617 Remission (n=164, n=69) | 29 | 13
  Day 729 LDAS (n=153, n=68) | 49 | 12
  Day 729 Remission (n=153, n=68) | 31 | 7
  Day 813 LDAS (n=139, n=58) | 43 | 16
  Day 813 Remission (n=139, n=58) | 26 | 6
  Day 897 LDAS (n=134, n=60) | 50 | 14
  Day 897 Remission (n=134, n=60) | 26 | 8
  Day 981 LDAS (n=121, n=49) | 47 | 14
  Day 981 Remission (n=121, n=49) | 28 | 7
  Day 1093 LDAS (n=134, n=56) | 50 | 15
  Day 1093 Remission (n=134, n=56) | 31 | 8
  Day 1261 LDAS (n=126, n=51) | 50 | 19
  Day 1261 Remission (n=126, n=51) | 25 | 9
  Day 1457 LDAS (n=115, n=50) | 46 | 14
  Day 1457 Remission (n=115, n=50) | 24 | 9
  Day 1625 LDAS (n=107, n=46) | 40 | 14
  Day 1625 Remission (n=107, n=46) | 28 | 11
  Day 1821 LDAS (n=103, n=45) | 38 | 12
  Day 1821 Remission (n=103, n=45) | 23 | 10

44. Secondary Outcome: OL; Mean Time-matched Baseline DAS28 (CRP) Over Time For Participants Treated in the OL
Description: The DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP levels, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Time-matched baseline values were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 209 | 98
units on a scale
  Day 15 cohort (n=206, n=95) | 6.52 (0.84) | 6.46 (0.81)
  Day 29 cohort (n=204, n=96) | 6.53 (0.86) | 6.46 (0.82)
  Day 57 cohort (n=207, n=97) | 6.51 (0.84) | 6.43 (0.81)
  Day 85 cohort (n=209, n=98) | 6.55 (0.84) | 6.45 (0.82)
  Day 113 cohort (n=199, n=93) | 6.55 (0.85) | 6.49 (0.80)
  Day 141 cohort (n=210, n=96) | 6.53 (0.85) | 6.43 (0.82)
  Day 169 cohort (n=205, n=96) | 6.54 (0.85) | 6.44 (0.81)
  Day 253 cohort (n=193, n=89) | 6.53 (0.86) | 6.44 (0.79)
  Day 365 cohort (n=192, n=93) | 6.51 (0.85) | 6.43 (0.83)
  Day 449 cohort (n=168, n=76) | 6.52 (0.86) | 6.42 (0.83)
  Day 533 cohort (n=162, n=73) | 6.52 (0.85) | 6.45 (0.78)
  Day 617 cohort (n=163, n=69) | 6.51 (0.82) | 6.49 (0.75)
  Day 729 cohort (n=151, n=68) | 6.50 (0.84) | 6.52 (0.76)
  Day 813 cohort (n=137, n=58) | 6.47 (0.83) | 6.56 (0.78)
  Day 897 cohort (n=132, n=60) | 6.43 (0.82) | 6.61 (0.73)
  Day 981 cohort (n=119, n=49) | 6.46 (0.84) | 6.56 (0.72)
  Day 1093 cohort (n=133, n=56) | 6.49 (0.81) | 6.53 (0.77)
  Day 1261 cohort (n=124, n=51) | 6.42 (0.83) | 6.50 (0.76)
  Day 1457 cohort (n=113, n=50) | 6.41 (0.83) | 6.54 (0.77)
  Day 1625 cohort (n=105, n=46) | 6.44 (0.85) | 6.50 (0.79)
  Day 1821 cohort (n=101, n=45) | 6.47 (0.82) | 6.54 (0.78)

45. Secondary Outcome: OL; Mean Time-matched Change From Baseline in DAS28 (CRP) Over Time For Participants Treated in the OL
Description: DAS28 is a continuous disease measure which is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, ESR or CRP, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (> 5.1), low disease activity (< 3.2) and remission (< 2.6). Time-matched mean change from baseline = Post-baseline value - time-matched baseline value, where the time-matched baseline value represents the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 15, 29, 57, 85, 113, 141, 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1261, 1457, 1625, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 209 | 98
units on a scale
  Day 15 cohort (n=206, n=95) | -0.74 (0.06) | -0.40 (0.08)
  Day 29 cohort (n=204, n=96) | -1.15 (0.07) | -0.72 (0.11)
  Day 57 cohort (n=207, n=97) | -1.59 (0.08) | -1.05 (0.12)
  Day 85 cohort (n=209, n=98) | -1.75 (0.08) | -0.88 (0.12)
  Day 113 cohort (n=199, n=93) | -1.92 (0.09) | -1.00 (0.13)
  Day 141 cohort (n=210, n=96) | -2.03 (0.09) | -1.05 (0.13)
  Day 169 cohort (n=205, n=96) | -2.00 (0.10) | -0.93 (0.12)
  Day 253 cohort (n=193, n=89) | -2.11 (0.09) | -2.03 (0.15)
  Day 365 cohort (n=192, n=93) | -2.33 (0.10) | -2.13 (0.15)
  Day 449 cohort (n=168, n=76) | -2.43 (0.11) | -2.49 (0.15)
  Day 533 cohort (n=162, n=73) | -2.57 (0.11) | -2.50 (0.16)
  Day 617 cohort (n=163, n=69) | -2.65 (0.10) | -2.58 (0.14)
  Day 729 cohort (n=151, n=68) | -2.66 (0.11) | -2.23 (0.17)
  Day 813 cohort (n=137, n=58) | -2.70 (0.12) | -2.40 (0.15)
  Day 897 cohort (n=132, n=60) | -2.73 (0.11) | -2.61 (0.16)
  Day 981 cohort (n=119, n=49) | -2.76 (0.13) | -2.66 (0.17)
  Day 1093 cohort (n=133, n=56) | -2.84 (0.12) | -2.62 (0.20)
  Day 1261 cohort (n=124, n=51) | -2.83 (0.12) | -2.85 (0.18)
  Day 1457 cohort (n=113, n=50) | -2.78 (0.13) | -2.78 (0.19)
  Day 1625 cohort (n=105, n=46) | -2.88 (0.13) | -2.80 (0.20)
  Day 1821 cohort (n=101, n=45) | -2.89 (0.14) | -2.98 (0.18)

46. Secondary Outcome: OL; Mean Time-matched Baseline DAS28 (ESR) Over Time For Participants Treated in the OL
Description: as for outcome 44
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 178 | 83
units on a scale
  Day 169 cohort (n=178, n=83) | 6.89 (1.00) | 6.83 (0.98)
  Day 253 cohort (n=163, n=75) | 6.87 (1.00) | 6.85 (1.01)
  Day 365 cohort (n=176, n=82) | 6.91 (1.01) | 6.80 (1.03)
  Day 449 cohort (n=152, n=70) | 6.94 (0.99) | 6.85 (0.97)
  Day 533 cohort (n=134, n=66) | 6.89 (1.02) | 6.81 (0.81)
  Day 617 cohort (n=143, n=59) | 6.86 (0.98) | 6.88 (0.82)
  Day 729 cohort (n=133, n=64) | 6.85 (1.01) | 6.86 (0.89)
  Day 813 cohort (n=120, n=52) | 6.84 (0.94) | 6.93 (0.93)
  Day 897 cohort (n=118, n=56) | 6.78 (0.96) | 6.93 (0.85)
  Day 981 cohort (n=119, n=50) | 6.85 (0.96) | 6.91 (0.84)
  Day 1093 cohort (n=111, n=50) | 6.84 (0.95) | 6.92 (0.88)
  Day 1261 cohort (n=107, n=50) | 6.77 (0.97) | 6.88 (0.87)
  Day 1457 cohort (n=94, n=45) | 6.80 (0.99) | 6.87 (0.89)
  Day 1625 cohort (n=89, n=41) | 6.81 (0.99) | 6.89 (0.90)
  Day 1821 cohort (n=87, n=42) | 6.85 (0.99) | 6.91 (0.91)

47. Secondary Outcome: OL; Mean Time-matched Change From Baseline in DAS28 (ESR) Over Time For Participants Treated in the OL
Description: as for outcome 45
Time Frame: BL, Days 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1261, 1457, 1625, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 178 | 83
units on a scale
  Day 169 cohort (n=178, n=83) | -2.05 (0.12) | -0.83 (0.14)
  Day 253 cohort (n=163, n=75) | -2.09 (0.11) | -2.00 (0.16)
  Day 365 cohort (n=176, n=82) | -2.31 (0.11) | -2.05 (0.17)
  Day 449 cohort (n=152, n=70) | -2.48 (0.12) | -2.53 (0.16)
  Day 533 cohort (n=134, n=66) | -2.48 (0.13) | -2.59 (0.16)
  Day 617 cohort (n=143, n=59) | -2.65 (0.12) | -2.60 (0.15)
  Day 729 cohort (n=133, n=64) | -2.65 (0.12) | -2.25 (0.16)
  Day 813 cohort (n=120, n=52) | -2.77 (0.13) | -2.43 (0.16)
  Day 897 cohort (n=118, n=56) | -2.65 (0.12) | -2.70 (0.17)
  Day 981 cohort (n=119, n=50) | -2.77 (0.13) | -2.59 (0.20)
  Day 1093 cohort (n=111, n=50) | -2.78 (0.14) | -2.56 (0.23)
  Day 1261 cohort (n=107, n=50) | -2.70 (0.15) | -2.56 (0.21)
  Day 1457 cohort (n=94, n=45) | -2.68 (0.15) | -2.58 (0.22)
  Day 1625 cohort (n=89, n=41) | -2.69 (0.15) | -2.64 (0.24)
  Day 1821 cohort (n=87, n=42) | -2.77 (0.15) | -2.73 (0.22)

48. Secondary Outcome: OL; Number of Participants Achieving HAQ Response Over Time In Participants Treated in the OL
Description: The HAQ disability index (HAQ DI) is a self-administered questionnaire composed of 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. The questions are evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. The HAQ disease index is a weighted sum of the scale scores, with a higher score indicating poorer function. Clinically meaningful HAQ response was defined as an improvement of at least 0.3 units from baseline in HAQ DI.
Time Frame: Days 15, 29, 57, 85, 113, 141, 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1261, 1457, 1625, and 1821
Population: Analysis was carried out on the intent-to-treat (ITT) population defined as all randomized subjects who received at least one dose of study medication. Two participants were unevaluable for response due to each missing 2 infusions of study drug. N=Number of Participants analyzed, n=number of participants with measurements at visit.
Measure: Number; unit: participants
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 209 | 98
participants
  Day 15 (n=209, n=96) | 59 | 16
  Day 29 (n=207, n=97) | 82 | 30
  Day 57 (n=209, n=98) | 101 | 34
  Day 85 (n=207, n=97) | 119 | 28
  Day 113 (n=202, n=96) | 113 | 30
  Day 141 (n=209, n=97) | 115 | 29
  Day 169 (n=207, n=98) | 115 | 31
  Day 253 (n=199, n=93) | 111 | 47
  Day 365 (n=182, n=87) | 128 | 49
  Day 449 (n=182, n=87) | 108 | 47
  Day 533 (n=165, n=78) | 99 | 44
  Day 617 (n=161, n=71) | 101 | 40
  Day 729 (n=154, n=74) | 101 | 46
  Day 813 (n=139, n=61) | 88 | 34
  Day 897 (n=132, n=62) | 87 | 37
  Day 981 (n=141, n=59) | 92 | 37
  Day 1093 (n=128, n=54) | 88 | 34
  Day 1261 (n=126, n=56) | 80 | 41
  Day 1457 (n=117, n=50) | 81 | 34
  Day 1625 (n=109, n=49) | 69 | 31
  Day 1821 (n=104, n=47) | 65 | 31

49. Secondary Outcome: OL; Mean Time-matched Baseline HAQ-DI and HAQ Component Scores Over Time For Participants Treated in the OL
Description: The HAQ DI is a self-administered questionnaire composed of 20 questions to assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip and common activities. Questions are evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. HAQ-DI is a weighted sum of the scale scores, with a higher score indicating poorer function. Time-matched baseline values were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 209 | 98
units on a scale
  Day 169 HAQ-DI (n=207, n=98) | 1.82 (0.54) | 1.79 (0.60)
  Day 169 Dressing and Grooming (n=209, n=98) | 1.65 (0.73) | 1.54 (0.69)
  Day 169 Arising (n=209, n=98) | 1.41 (0.72) | 1.44 (0.73)
  Day 169 Eating (n=209, n=98) | 1.75 (0.84) | 1.80 (0.87)
  Day 169 Walking (n=208, n=96) | 1.57 (0.71) | 1.51 (0.75)
  Day 169 Hygiene (n=208, n=98) | 2.14 (0.88) | 2.21 (0.86)
  Day 169 Reaching (n=208, n=98) | 2.04 (0.79) | 1.97 (0.87)
  Day 169 Gripping (n=207, n=98) | 1.95 (0.53) | 1.92 (0.62)
  Day 169 Activities (n=208, n=98) | 2.01 (0.77) | 1.96 (0.86)
  Day 365 HAQ-DI (n=199, n=97) | 1.80 (0.56) | 1.80 (0.60)
  Day 365 Dressing and Grooming (n=201, n=97) | 1.62 (0.74) | 1.55 (0.69)
  Day 365 Arising (n=201, n=97) | 1.39 (0.71) | 1.45 (0.74)
  Day 365 Eating (n=201, n=97) | 1.73 (0.84) | 1.80 (0.87)
  Day 365 Walking (n=199, n=95) | 1.55 (0.73) | 1.51 (0.76)
  Day 365 Hygiene (n=201, n=97) | 2.14 (0.89) | 2.22 (0.87)
  Day 365 Reaching (n=201, n=97) | 2.03 (0.81) | 1.98 (0.97)
  Day 365 Gripping (n=200, n=97) | 1.94 (0.55) | 1.92 (0.62)
  Day 365 Activities (n=200, n=97) | 2.02 (0.80) | 1.96 (0.85)
  Day 729 HAQ-DI (n=154, n=74) | 1.77 (0.57) | 1.79 (0.59)
  Day 729 Dressing and Grooming (n=156, n=74) | 1.62 (0.74) | 1.54 (0.67)
  Day 729 Arising (n=156, n=74) | 1.37 (0.72) | 1.43 (0.70)
  Day 729 Eating (n=156, n=74) | 1.69 (0.86) | 1.81 (0.84)
  Day 729 Walking (n=156, n=72) | 1.53 (0.74) | 1.47 (0.73)
  Day 729 Hygiene (n=154, n=74) | 2.07 (0.91) | 2.23 (0.88)
  Day 729 Reaching (n=154, n=74) | 1.98 (0.83) | 2.03 (0.83)
  Day 729 Gripping (n=154, n=74) | 1.94 (0.55) | 1.88 (0.57)
  Day 729 Activities (n=154, n=74) | 2.01 (0.80) | 1.93 (0.85)
  Day 1093 HAQ-DI (n=128, n=54) | 1.78 (0.57) | 1.81 (0.54)
  Day 1093 Dressing and Grooming (n=129, n=54) | 1.62 (0.75) | 1.59 (0.57)
  Day 1093 Arising (n=129, n=54) | 1.38 (0.72) | 1.44 (0.72)
  Day 1093 Eating (n=129, n=54) | 1.68 (0.84) | 1.81 (0.80)
  Day 1093 Walking (n=129, n=54) | 1.55 (0.73) | 1.43 (0.69)
  Day 1093 Hygiene (n=135, n=59) | 2.04 (0.91) | 2.25 (0.86)
  Day 1093 Reaching (n=135, n=59) | 1.95 (0.83) | 2.14 (0.78)
  Day 1093 Gripping (n=135, n=59) | 1.95 (0.52) | 1.93 (0.49)
  Day 1093 Activities (n=135, n=59) | 1.96 (0.78) | 1.98 (0.80)
  Day 1457 HAQ-DI (n=117, n=50) | 1.75 (0.58) | 1.87 (0.54)
  Day 1457 Dressing and Grooming (n=117, n=50) | 1.64 (0.74) | 1.64 (0.56)
  Day 1457 Arising (n=117, n=50) | 1.35 (0.71) | 1.44 (0.73)
  Day 1457 Eating (n=117, n=50) | 1.67 (0.85) | 1.92 (0.85)
  Day 1457 Walking (n=117, n=50) | 1.50 (0.71) | 1.48 (0.71)
  Day 1457 Hygiene (n=118, n=50) | 2.06 (0.89) | 2.32 (0.82)
  Day 1457 Reaching (n=118, n=50) | 1.97 (0.83) | 2.12 (0.80)
  Day 1457 Gripping (n=118, n=50) | 1.93 (0.55) | 1.98 (0.43)
  Day 1457 Activities (n=118, n=50) | 1.92 (0.81) | 2.02 (0.82)
  Day 1821 HAQ-DI (n=104, n=47) | 1.75 (0.61) | 1.84 (0.57)
  Day 1821 Dressing and Grooming (n=105, n=47) | 1.65 (0.77) | 1.62 (0.57)
  Day 1821 Arising (n=105, n=47) | 1.38 (0.73) | 1.43 (0.74)
  Day 1821 Eating (n=105, n=47) | 1.62 (0.86) | 1.89 (0.89)
  Day 1821 Walking (n=103, n=47) | 1.51 (0.68) | 1.45 (0.72)
  Day 1821 Hygiene (n=104, n=47) | 2.02 (0.90) | 2.26 (0.85)
  Day 1821 Reaching (n=104, n=47) | 1.94 (0.85) | 2.11 (0.81)
  Day 1821 Gripping (n=104, n=47) | 1.93 (0.60) | 1.94 (0.53)
  Day 1821 Activities (n=104, n=47) | 1.93 (0.80) | 2.00 (0.86)

50. Secondary Outcome: OL; Mean Time-matched Change From Baseline in HAQ-DI and HAQ Component Scores For Participants Treated in the OL
Description: HAQ-DI is a self-administered questionnaire composed of 20 questions to assess physical functions in 8 domains:dressing, arising, eating, walking, hygiene, reach, grip and common activities. Questions evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. HAQ-DI=weighted sum of the scale scores. Higher score indicates poorer function.Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit
Time Frame: BL, Days 169, 253, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1261, 1457, 1625, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- OL: ABA: Participants with active RA who met the inclusion/exclusion criteria for this study were randomized to receive abatacept on a background of DMARDs. Participants must have been treated with anti-TNF therapy for at least 3 months and designated as anti-TNF therapy failures due to inadequate efficacy. Participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram. Study medication was administered on Days 1, 15, 29 and every 28 days thereafter for a total of 7 doses. Each dose was infused intravenously over approximately 30 minutes.
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 209 | 98
units on a scale
  Day 169 HAQ-DI (n=207, n=98) | -0.51 (0.04) | -0.16 (0.04)
  Day 169 Dressing and Grooming (n=209, n=98) | -0.60 (0.06) | -0.26 (0.07)
  Day 169 Arising (n=209, n=98) | -0.61 (0.05) | -0.31 (0.07)
  Day 169 Eating (n=209, n=98) | -0.53 (0.06) | -0.09 (0.06)
  Day 169 Walking (n=208, n=96) | -0.52 (0.05) | -0.23 (0.07)
  Day 169 Hygiene (n=208, n=98) | -0.28 (0.05) | -0.08 (0.07)
  Day 169 Reaching (n=208, n=98) | -0.55 (0.06) | -0.11 (0.06)
  Day 169 Gripping (n=207, n=98) | -0.46 (0.06) | -0.14 (0.06)
  Day 169 Activities (n=208, n=98) | -0.50 (0.06) | -0.09 (0.06)
  Day 365 HAQ-DI (n=199, n=97) | -0.52 (0.04) | -0.40 (0.05)
  Day 365 Dressing and Grooming (n=201, n=97) | -0.58 (0.06) | -0.44 (0.08)
  Day 365 Arising (n=201, n=97) | -0.50 (0.06) | -0.55 (0.07)
  Day 365 Eating (n=201, n=97) | -0.57 (0.06) | -0.47 (0.08)
  Day 365 Walking (n=199, n=95) | -0.50 (0.06) | -0.55 (0.08)
  Day 365 Hygiene (n=201, n=97) | -0.36 (0.06) | -0.28 (0.08)
  Day 365 Reaching (n=201, n=97) | -0.59 (0.06) | -0.33 (0.09)
  Day 365 Gripping (n=200, n=97) | -0.55 (0.06) | -0.28 (0.07)
  Day 365 Activities (n=200, n=97) | -0.51 (0.06) | -0.34 (0.08)
  Day 729 HAQ-DI (n=154, n=74) | -0.62 (0.05) | -0.50 (0.07)
  Day 729 Dressing and Grooming (n=156, n=74) | -0.74 (0.07) | -0.59 (0.10)
  Day 729 Arising (n=156, n=74) | -0.62 (0.06) | -0.64 (0.08)
  Day 729 Eating (n=156, n=74) | -0.69 (0.07) | -0.54 (0.09)
  Day 729 Walking (n=156, n=72) | -0.59 (0.07) | -0.49 (0.10)
  Day 729 Hygiene (n=154, n=74) | -0.35 (0.07) | -0.36 (0.11)
  Day 729 Reaching (n=154, n=74) | -0.64 (0.07) | -0.51 (0.10)
  Day 729 Gripping (n=154, n=74) | -0.62 (0.08) | -0.43 (0.09)
  Day 729 Activities (n=154, n=74) | -0.62 (0.06) | -0.46 (0.11)
  Day 1093 HAQ-DI (n=128, n=54) | -0.65 (0.05) | -0.51 (0.07)
  Day 1093 Dressing and Grooming (n=129, n=54) | -0.74 (0.07) | -0.65 (0.11)
  Day 1093 Arising (n=129, n=54) | -0.67 (0.07) | -0.72 (0.10)
  Day 1093 Eating (n=129, n=54) | -0.71 (0.07) | -0.57 (0.10)
  Day 1093 Walking (n=129, n=54) | -0.64 (0.08) | -0.52 (0.11)
  Day 1093 Hygiene (n=135, n=59) | -0.36 (0.07) | -0.37 (0.13)
  Day 1093 Reaching (n=135, n=59) | -0.63 (0.07) | -0.59 (0.10)
  Day 1093 Gripping (n=135, n=59) | -0.69 (0.08) | -0.31 (0.08)
  Day 1093 Activities (n=135, n=59) | -0.64 (0.07) | -0.54 (0.10)
  Day 1457 HAQ-DI (n=117, n=50) | -0.58 (0.05) | -0.62 (0.09)
  Day 1457 Dressing and Grooming (n=117, n=50) | -0.74 (0.08) | -0.76 (0.12)
  Day 1457 Arising (n=117, n=50) | -0.60 (0.07) | -0.74 (0.13)
  Day 1457 Eating (n=117, n=50) | -0.64 (0.08) | -0.70 (0.14)
  Day 1457 Walking (n=117, n=50) | -0.50 (0.08) | -0.64 (0.13)
  Day 1457 Hygiene (n=118, n=50) | -0.29 (0.08) | -0.54 (0.14)
  Day 1457 Reaching (n=118, n=50) | -0.68 (0.07) | -0.60 (0.13)
  Day 1457 Gripping (n=118, n=50) | -0.55 (0.08) | -0.38 (0.11)
  Day 1457 Activities (n=118, n=50) | -0.59 (0.08) | -0.56 (0.11)
  Day 1821 HAQ-DI (n=104, n=47) | -0.57 (0.06) | -0.66 (0.09)
  Day 1821 Dressing and Grooming (n=105, n=47) | -0.75 (0.08) | -0.83 (0.12)
  Day 1821 Arising (n=105, n=47) | -0.59 (0.08) | -0.79 (0.12)
  Day 1821 Eating (n=105, n=47) | -0.54 (0.08) | -0.87 (0.12)
  Day 1821 Walking (n=103, n=47) | -0.54 (0.09) | -0.57 (0.12)
  Day 1821 Hygiene (n=104, n=47) | -0.27 (0.09) | -0.57 (0.16)
  Day 1821 Reaching (n=104, n=47) | -0.68 (0.09) | -0.62 (0.10)
  Day 1821 Gripping (n=104, n=47) | -0.58 (0.09) | -0.40 (0.11)
  Day 1821 Activities (n=104, n=47) | -0.59 (0.08) | -0.64 (0.12)

51. Secondary Outcome: OL; Mean Time-matched Baseline Levels of Rheumatoid Factor (RF) Over Time For Participants Treated in the OL
Description: RF is an autoantibody most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process. Time-matched baseline levels of RF were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 191 | 95
IU/ml
  Day 169 cohort (n=191, n=95) | 262.4 (487.9) | 264.8 (430.4)
  Day 365 cohort (n=189, n=92) | 275.5 (505.4) | 270.4 (435.9)
  Day 729 cohort (n=150, n=71) | 276.8 (513.1) | 301.5 (476.4)
  Day 1093 cohort (n=123, n=57) | 234.6 (404.4) | 328.9 (509.8)
  Day 1457 cohort (n=106, n=46) | 247.8 (368.0) | 331.3 (552.9)
  Day 1821 cohort (n=97, n=45) | 214.8 (348.4) | 318.4 (552.3)

52. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Levels of RF Over Time For Participants Treated in the OL
Description: RF is an autoantibody most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes which contribute to the disease process. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1261, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: IU/ml
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 191 | 95
IU/ml
  Day 169 cohort (n=191, n=95) | -80.4 (20.17) | -25.1 (18.54)
  Day 365 cohort (n=189, n=92) | -50.0 (28.64) | -69.6 (24.58)
  Day 729 cohort (n=150, n=71) | -30.2 (40.77) | -82.8 (41.86)
  Day 1093 cohort (n=123, n=57) | -6.70 (46.76) | -86.5 (65.61)
  Day 1457 cohort (n=106, n=46) | 6.79 (42.12) | -68.1 (86.80)
  Day 1821 cohort (n=97, n=45) | -10.7 (32.57) | -103.0 (83.56)

53. Secondary Outcome: OL; Mean Time-matched Baseline Levels of C-Reactive Protein (CRP) Over Time For Participants Treated in the OL
Description: CRP is an acute phase reactant protein that is a clinical marker for Rheumatoid Arthritis (RA). Time-matched baseline levels of CRP were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 210 | 99
mg/dL
  Day 169 cohort (n=210, n=99) | 46.00 (38.77) | 33.34 (31.13)
  Day 365 cohort (n=196, n=95) | 45.62 (39.31) | 34.05 (31.55)
  Day 729 cohort (n=158, n=71) | 45.61 (39.11) | 34.60 (30.69)
  Day 1093 cohort (n=139, n=59) | 43.20 (37.17) | 35.07 (29.95)
  Day 1457 cohort (n=125, n=52) | 41.98 (36.52) | 35.30 (30.87)
  Day 1821 cohort (n=108, n=46) | 41.23 (35.71) | 34.83 (28.26)

54. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Levels of CRP Over Time For Participants Treated in the OL
Description: CRP is an acute phase reactant protein that is a clinical marker for RA. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1261, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 210 | 99
mg/dL
  Day 169 cohort (n=210, n=99) | -25.3 (2.70) | -0.36 (3.24)
  Day 365 cohort (n=196, n=95) | -29.1 (2.72) | -16.8 (3.07)
  Day 729 cohort (n=158, n=71) | -29.4 (3.30) | -10.8 (4.68)
  Day 1093 cohort (n=139, n=59) | -31.8 (3.08) | -18.8 (3.23)
  Day 1457 cohort (n=125, n=52) | -30.1 (3.30) | -22.8 (4.86)
  Day 1821 cohort (n=108, n=46) | -30.1 (3.47) | -23.2 (4.33)

55. Secondary Outcome: OL; Mean Time-matched Baseline Erythrocyte Sedimentation Rate (ESR) Over Time For Participants Treated in the OL
Description: ESR, also called a sedimentation rate or Biernacki Reaction, is the rate at which red blood cells sediment in a period of 1 hour. It is a common hematology test that is a non-specific measure of inflammation. Time-matched baseline levels of ESR were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 174 | 81
mm/hr
  Day 169 cohort (n=174, n=81) | 50.60 (28.06) | 44.40 (26.64)
  Day 365 cohort (n=171, n=81) | 50.51 (28.61) | 44.10 (26.41)
  Day 729 cohort (n=135, n=67) | 50.53 (28.52) | 42.06 (23.77)
  Day 1093 cohort (n=113, n=53) | 49.03 (26.11) | 43.36 (24.42)
  Day 1457 cohort (n=99, n=45) | 50.04 (26.91) | 42.64 (25.76)
  Day 1821 cohort (n=90, n=43) | 50.32 (26.41) | 43.02 (24.96)

56. Secondary Outcome: OL; Mean Time-matched Change From Baseline in ESR Over Time For Participants Treated in the OL
Description: ESR, also called a sedimentation rate or Biernacki Reaction, is the rate at which red blood cells sediment in a period of 1 hour. It is a common hematology test that is a non-specific measure of inflammation. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1261, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mm/hr
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 174 | 81
mm/hr
  Day 169 cohort (n=174, n=81) | -18.0 (1.89) | -0.44 (2.60)
  Day 365 cohort (n=171, n=81) | -18.8 (1.97) | -10.1 (2.50)
  Day 729 cohort (n=135, n=67) | -20.2 (2.48) | -6.25 (3.15)
  Day 1093 cohort (n=113, n=53) | -19.9 (2.54) | -10.6 (3.60)
  Day 1457 cohort (n=99, n=45) | -20.5 (2.56) | -9.80 (4.44)
  Day 1821 cohort (n=90, n=43) | -19.5 (2.79) | -9.49 (4.45)

57. Secondary Outcome: OL; Mean Time-matched Baseline Levels of Soluble Interleukin 2 Receptor (sIL-2R) Over Time For Participants Treated in the OL
Description: IL-2 is a proinflammatory cytokine, and the soluble form of its receptor (IL-2R) is a marker for inflammation. Time-matched baseline levels of IL-2R were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 198 | 91
pg/ml
  Day 169 cohort (n=198, n=91) | 1879.0 (909.3) | 1805.0 (922.9)
  Day 365 cohort (n=183, n=88) | 1851.0 (762.5) | 1800.0 (941.5)
  Day 729 cohort (n=135, n=66) | 1942.0 (971.5) | 1708.0 (864.9)
  Day 1093 cohort (n=72, n=36) | 1813.0 (781.8) | 1827.0 (974.2)

58. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Levels of sIL-2R Over Time For Participants Treated in the OL
Description: IL-2 is a proinflammatory cytokine, and the soluble form of its receptor (IL-2R) is a marker for inflammation. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1261, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 198 | 91
pg/ml
  Day 169 cohort (n=198, n=91) | -590.0 (41.75) | -19.6 (73.21)
  Day 365 cohort (n=183, n=88) | -522.0 (50.84) | -424.0 (71.42)
  Day 729 cohort (n=135, n=66) | -836.0 (58.94) | -483.0 (101.6)
  Day 1093 cohort (n=72, n=36) | -761.0 (92.88) | -794.0 (136.1)

59. Secondary Outcome: OL; Mean Time-matched Baseline SF-36 PCS and MCS Over Time For Participants Treated in OL
Description: SF-36 measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores:PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Time-matched baseline values were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 204 | 98
units on a scale
  Day 169 cohort (n=204, n=98): PCS | 27.52 (6.65) | 28.07 (6.86)
  Day 365 cohort (n=198, n=96): PCS | 27.70 (6.76) | 27.92 (6.83)
  Day 729 cohort (n=155, n=73): PCS | 27.81 (6.69) | 28.65 (6.80)
  Day 1093 cohort (n=130, n=58): PCS | 27.92 (6.86) | 28.25 (6.72)
  Day 1457 cohort (n=114, n=50): PCS | 28.31 (6.85) | 28.06 (6.85)
  Day 1821 cohort (n=103, n=47): PCS | 28.48 (6.72) | 28.27 (6.97)
  Day 169 cohort (n=204, n=98): MCS | 41.75 (12.53) | 43.62 (12.12)
  Day 365 cohort (n=198, n=96): MCS | 41.54 (12.69) | 43.96 (11.98)
  Day 729 cohort (n=155, n=73): MCS | 42.23 (12.86) | 42.42 (11.89)
  Day 1093 cohort (n=130, n=58): MCS | 43.29 (12.25) | 42.13 (11.75)
  Day 1457 cohort (n=114, n=50): MCS | 43.38 (12.20) | 41.95 (11.67)
  Day 1821 cohort (n=103, n=47): MCS | 41.74 (12.82) | 42.70 (11.64)

60. Secondary Outcome: OL; Mean Time-matched Change From Baseline in SF-36 PCS and MCS Over Time For Participants Treated in OL
Description: SF-36 measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 204 | 98
units on a scale
  Day 169 cohort (n=204, n=98): PCS | 7.46 (0.69) | 1.90 (0.77)
  Day 365 cohort (n=198, n=96): PCS | 8.30 (0.74) | 6.21 (0.94)
  Day 729 cohort (n=155, n=73): PCS | 10.28 (0.78) | 6.79 (1.16)
  Day 1093 cohort (n=130, n=58): PCS | 10.30 (0.90) | 8.61 (1.34)
  Day 1457 cohort (n=114, n=50): PCS | 8.71 (0.93) | 8.51 (1.39)
  Day 1821 cohort (n=103, n=47): PCS | 9.32 (1.06) | 9.35 (1.52)
  Day 169 cohort (n=204, n=98): MCS | 5.83 (0.83) | 2.16 (0.91)
  Day 365 cohort (n=198, n=96): MCS | 5.18 (0.79) | 5.32 (1.07)
  Day 729 cohort (n=155, n=73): MCS | 6.08 (0.92) | 8.61 (1.42)
  Day 1093 cohort (n=130, n=58): MCS | 5.68 (1.05) | 9.14 (1.72)
  Day 1457 cohort (n=114, n=50): MCS | 5.41 (1.12) | 7.93 (1.77)
  Day 1821 cohort (n=103, n=47): MCS | 6.42 (1.24) | 10.37 (1.75)

61. Secondary Outcome: OL; Mean Time-matched Baseline Physical Function Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=208, n=98): Physical Function | 26.22 (8.75) | 26.60 (8.65)
  Day 365 cohort (n=200, n=96): Physical Function | 26.37 (8.88) | 26.49 (8.62)
  Day 729 cohort (n=156, n=74): Physical Function | 27.03 (9.03) | 26.66 (8.37)
  Day 1093 cohort (n=133, n=59): Physical Function | 27.06 (9.03) | 25.66 (7.99)
  Day 1457 cohort (n=118, n=50): Physical Function | 27.54 (9.15) | 25.41 (8.08)
  Day 1821 cohort (n=104, n=47): Physical Function | 27.86 (9.65) | 25.61 (8.45)

62. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Physical Function Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=208, n=98): Physical Function | 5.75 (0.74) | 1.82 (0.84)
  Day 365 cohort (n=200, n=96): Physical Function | 7.14 (0.79) | 4.80 (0.97)
  Day 729 cohort (n=156, n=74): Physical Function | 7.61 (0.90) | 7.38 (1.09)
  Day 1093 cohort (n=133, n=59): Physical Function | 8.24 (1.00) | 9.68 (1.26)
  Day 1457 cohort (n=118, n=50): Physical Function | 6.36 (1.06) | 8.98 (1.32)
  Day 1821 cohort (n=104, n=47): Physical Function | 7.34 (1.21) | 8.57 (1.63)

63. Secondary Outcome: OL; Mean Time-matched Baseline Role-Physical Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=210, n=98): Role-Physical | 30.50 (6.20) | 32.36 (7.36)
  Day 365 cohort (n=203, n=97): Role-Physical | 30.49 (6.24) | 32.40 (7.38)
  Day 729 cohort (n=156, n=74): Role-Physical | 30.48 (6.02) | 32.45 (7.08)
  Day 1093 cohort (n=135, n=59): Role-Physical | 30.71 (6.42) | 31.91 (6.98)
  Day 1457 cohort (n=117, n=50): Role-Physical | 31.20 (6.81) | 31.91 (7.02)
  Day 1821 cohort (n=106, n=47): Role-Physical | 30.93 (6.63) | 32.47 (7.58)

64. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Role-Physical Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=210, n=98): Role-Physical | 7.82 (0.80) | 1.30 (0.99)
  Day 365 cohort (n=203, n=97): Role-Physical | 7.78 (0.85) | 6.49 (1.25)
  Day 729 cohort (n=156, n=74): Role-Physical | 10.76 (0.97) | 6.59 (1.42)
  Day 1093 cohort (n=135, n=59): Role-Physical | 10.27 (1.10) | 8.91 (1.58)
  Day 1457 cohort (n=117, n=50): Role-Physical | 9.09 (1.11) | 7.64 (1.75)
  Day 1821 cohort (n=106, n=47): Role-Physical | 9.05 (1.28) | 9.93 (1.87)

65. Secondary Outcome: OL; Mean Time-matched Baseline Bodily Pain Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=209, n=98): Bodily Pain | 30.76 (6.77) | 31.90 (6.55)
  Day 365 cohort (n=202, n=97): Bodily Pain | 30.75 (6.80) | 31.84 (6.56)
  Day 729 cohort (n=156, n=74): Bodily Pain | 31.00 (6.77) | 31.98 (6.65)
  Day 1093 cohort (n=135, n=59): Bodily Pain | 31.41 (6.86) | 31.71 (6.32)
  Day 1457 cohort (n=117, n=50): Bodily Pain | 31.73 (6.85) | 31.38 (6.31)
  Day 1821 cohort (n=106, n=47): Bodily Pain | 31.60 (7.07) | 31.78 (6.67)

66. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Bodily Pain Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=209, n=98): Bodily Pain | 9.59 (0.72) | 3.32 (0.78)
  Day 365 cohort (n=202, n=97): Bodily Pain | 10.25 (0.73) | 9.55 (0.98)
  Day 729 cohort (n=156, n=74): Bodily Pain | 12.36 (0.80) | 10.29 (1.23)
  Day 1093 cohort (n=135, n=59): Bodily Pain | 12.33 (0.95) | 11.34 (1.45)
  Day 1457 cohort (n=117, n=50): Bodily Pain | 10.79 (0.91) | 11.52 (1.60)
  Day 1821 cohort (n=106, n=47): Bodily Pain | 11.83 (1.13) | 14.33 (1.43)

67. Secondary Outcome: OL; Mean Time-matched Baseline General Health Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98): General Health | 35.28 (9.49) | 35.52 (8.76)
  Day 365 cohort (n=204, n=97): General Health | 35.50 (9.55) | 35.48 (8.76)
  Day 729 cohort (n=157, n=74): General Health | 35.49 (9.79) | 35.48 (8.98)
  Day 1093 cohort (n=136, n=59): General Health | 36.21 (9.79) | 35.78 (8.79)
  Day 1457 cohort (n=119, n=50): General Health | 36.21 (9.99) | 35.92 (8.92)
  Day 1821 cohort (n=106, n=47): General Health | 35.50 (10.1) | 36.14 (9.02)

68. Secondary Outcome: OL; Mean Time-matched Change From Baseline in General Health Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98): General Health | 4.48 (0.59) | 1.09 (0.82)
  Day 365 cohort (n=204, n=97): General Health | 4.36 (0.60) | 4.04 (0.84)
  Day 729 cohort (n=157, n=74): General Health | 6.43 (0.67) | 5.85 (0.98)
  Day 1093 cohort (n=136, n=59): General Health | 6.05 (0.71) | 5.92 (1.35)
  Day 1457 cohort (n=119, n=50): General Health | 5.29 (0.82) | 5.60 (1.41)
  Day 1821 cohort (n=106, n=47): General Health | 5.75 (0.81) | 6.92 (1.46)

69. Secondary Outcome: OL; Mean Time-matched Baseline Vitality Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98): Vitality | 35.06 (8.82) | 36.51 (9.15)
  Day 365 cohort (n=204, n=97): Vitality | 35.09 (8.73) | 36.65 (9.09)
  Day 729 cohort (n=157, n=74): Vitality | 35.45 (9.00) | 36.50 (8.95)
  Day 1093 cohort (n=136, n=59): Vitality | 35.74 (9.06) | 36.53 (8.23)
  Day 1457 cohort (n=118, n=50): Vitality | 35.94 (8.99) | 35.83 (8.18)
  Day 1821 cohort (n=105, n=47): Vitality | 35.01 (8.54) | 36.35 (8.47)

70. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Vitality Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98): Vitality | 7.80 (0.75) | 2.89 (0.87)
  Day 365 cohort (n=204, n=97): Vitality | 8.00 (0.76) | 6.69 (0.98)
  Day 729 cohort (n=157, n=74): Vitality | 8.49 (0.83) | 7.52 (1.20)
  Day 1093 cohort (n=136, n=59): Vitality | 8.23 (0.96) | 8.61 (1.63)
  Day 1457 cohort (n=118, n=50): Vitality | 7.62 (0.96) | 8.08 (1.76)
  Day 1821 cohort (n=105, n=47): Vitality | 8.51 (1.05) | 9.82 (1.69)

71. Secondary Outcome: OL; Mean Time-matched Baseline Social Functioning Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=211, n=98): Social Functioning | 33.31 (11.01) | 34.37 (11.42)
  Day 365 cohort (n=204, n=97): Social Functioning | 33.59 (11.01) | 34.30 (11.46)
  Day 729 cohort (n=157, n=74): Social Functioning | 33.87 (11.22) | 34.32 (11.29)
  Day 1093 cohort (n=136, n=59): Social Functioning | 34.43 (10.86) | 34.14 (11.46)
  Day 1457 cohort (n=119, n=50): Social Functioning | 35.20 (11.12) | 33.36 (11.60)
  Day 1821 cohort (n=106, n=47): Social Functioning | 34.91 (11.62) | 34.15 (11.88)

72. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Social Functioning Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=211, n=98): Social Functioning | 8.36 (0.85) | 2.99 (1.12)
  Day 365 cohort (n=204, n=97): Social Functioning | 8.17 (0.85) | 7.22 (1.28)
  Day 729 cohort (n=157, n=74): Social Functioning | 9.89 (0.96) | 9.10 (1.48)
  Day 1093 cohort (n=136, n=59): Social Functioning | 10.46 (1.05) | 10.49 (1.54)
  Day 1457 cohort (n=119, n=50): Social Functioning | 8.62 (1.08) | 11.83 (1.92)
  Day 1821 cohort (n=106, n=47): Social Functioning | 9.17 (1.16) | 12.24 (1.79)

73. Secondary Outcome: OL; Mean Time-matched Baseline Role-Emotional Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=210, n=98): Role-Emotional | 35.73 (13.69) | 37.60 (14.00)
  Day 365 cohort (n=203, n=97): Role-Emotional | 35.93 (13.73) | 37.75 (14.00)
  Day 729 cohort (n=156, n=73): Role-Emotional | 36.09 (13.65) | 35.86 (13.45)
  Day 1093 cohort (n=134, n=58): Role-Emotional | 36.87 (13.82) | 35.54 (13.54)
  Day 1457 cohort (n=117, n=50): Role-Emotional | 37.06 (13.58) | 36.17 (13.74)
  Day 1821 cohort (n=106, n=47): Role-Emotional | 36.26 (13.80) | 36.29 (13.65)

74. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Role-Emotional Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=210, n=98): Role-Emotional | 7.17 (1.11) | 1.83 (1.40)
  Day 365 cohort (n=203, n=97): Role-Emotional | 5.47 (1.04) | 6.52 (1.58)
  Day 729 cohort (n=156, n=73): Role-Emotional | 7.29 (1.18) | 10.39 (1.94)
  Day 1093 cohort (n=134, n=58): Role-Emotional | 6.88 (1.36) | 11.62 (2.28)
  Day 1457 cohort (n=117, n=50): Role-Emotional | 6.66 (1.49) | 6.32 (2.39)
  Day 1821 cohort (n=106, n=47): Role-Emotional | 7.26 (1.55) | 12.10 (2.35)

75. Secondary Outcome: OL; Mean Time-matched Baseline Mental Health Score Over Time For Participants Treated in the OL
Description: as for outcome 59
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98): Mental Health | 40.96 (13.07) | 43.47 (11.34)
  Day 365 cohort (n=204, n=97): Mental Health | 41.11 (13.06) | 43.53 (11.37)
  Day 729 cohort (n=157, n=73): Mental Health | 41.85 (13.38) | 42.69 (10.81)
  Day 1093 cohort (n=136, n=59): Mental Health | 42.68 (12.58) | 41.85 (10.54)
  Day 1457 cohort (n=118, n=50): Mental Health | 42.52 (12.74) | 41.44 (10.62)
  Day 1821 cohort (n=105, n=47): Mental Health | 41.36 (13.05) | 42.50 (10.36)

76. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Mental Health Score Over Time For Participants Treated in the OL
Description: as for outcome 60
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98): Mental Health | 4.42 (0.71) | 1.65 (0.83)
  Day 365 cohort (n=204, n=97): Mental Health | 4.53 (0.73) | 4.29 (0.93)
  Day 729 cohort (n=157, n=73): Mental Health . | 5.54 (0.84) | 7.19 (1.29)
  Day 1093 cohort (n=136, n=59): Mental Health | 5.24 (0.95) | 7.69 (1.45)
  Day 1457 cohort (n=118, n=50): Mental Health | 4.60 (0.89) | 8.91 (1.41)
  Day 1821 cohort (n=105, n=47): Mental Health | 5.31 (1.08) | 8.66 (1.53)

77. Secondary Outcome: OL; Mean Time-matched Baseline Medical Outcomes Study Sleep Module (MOS-sleep) Score Over Time For Participants Treated in the OL
Description: The validated 12-it3em Medical Outcomes Study sleep questionnaire (MOS-sleep) was used to measure sleep quality. An overall Sleep Problem Index (SPI) was generated as a summary measure of different types of sleep problems (sleep disturbance, sleep quantity, sleep adequacy, etc.). The score ranges from 0 to 100 with a higher score reflecting more severe problems with sleep. The mean score of the SPI in a population with chronic problems is 29.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98) | 49.18 (18.10) | 45.49 (17.72)
  Day 365 cohort (n=204, n=97) | 48.87 (19.09) | 45.54 (17.86)
  Day 729 cohort (n=157, n=74) | 48.62 (18.12) | 45.36 (17.26)
  Day 1093 cohort (n=136, n=59) | 48.01 (17.86) | 46.44 (17.28)
  Day 1457 cohort (n=119, n=50) | 46.71 (17.97) | 47.14 (18.47)
  Day 1821 cohort (n=106, n=47) | 47.49 (17.27) | 45.09 (17.90)

78. Secondary Outcome: OL; Mean Time-matched Change From Baseline in MOS-Sleep Score Over Time For Participants Treated in the OL
Description: The validated 12-it3em Medical Outcomes Study sleep questionnaire (MOS-sleep) was used to measure sleep quality. An overall Sleep Problem Index (SPI) was generated as a summary measure of different types of sleep problems (sleep disturbance, sleep quantity, sleep adequacy, etc.). The score ranges from 0 to 100 with a higher score reflecting more severe problems with sleep. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 208 | 98
units on a scale
  Day 169 cohort (n=212, n=98) | -11.1 (1.10) | -4.31 (1.59)
  Day 365 cohort (n=204, n=97) | -11.2 (1.33) | -10.4 (1.82)
  Day 729 cohort (n=157, n=74) | -12.5 (1.38) | -11.9 (2.06)
  Day 1093 cohort (n=136, n=59) | -12.9 (1.47) | -16.1 (2.53)
  Day 1457 cohort (n=119, n=50) | -9.86 (1.56) | -11.9 (2.92)
  Day 1821 cohort (n=106, n=47) | -11.7 (1.55) | -15.9 (2.84)

79. Secondary Outcome: OL; Mean Time-matched Baseline Fatigue Visual Analog Score (VAS) Over Time For Participants Treated in the OL
Description: Fatigue severity was assessed on the VAS 100 mm where 0= no fatigue to 100 = the worst fatigue imaginable. Time-matched baseline values were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 212 | 98
units on a scale
  Day 169 cohort (n=212, n=98) | 73.73 (19.84) | 71.24 (20.27)
  Day 365 cohort (n=204, n=97) | 73.54 (20.00) | 70.78 (20.13)
  Day 729 cohort (n=157, n=74) | 73.75 (19.18) | 69.59 (20.74)
  Day 1093 cohort (n=135, n=59) | 73.21 (19.93) | 70.00 (21.00)
  Day 1457 cohort (n=119, n=50) | 72.15 (19.73) | 71.14 (19.57)
  Day 1821 cohort (n=106, n=47) | 72.36 (20.51) | 69.68 (20.08)

80. Secondary Outcome: OL; Mean Time-matched Change From Baseline in Fatigue VAS Over Time For Participants Treated in the OL
Description: Fatigue severity was assessed on the VAS 100 mm where 0= no fatigue to 100 = the worst fatigue imaginable. Change from BL = Post-BL value - time-matched BL value, where the time-matched BL value represents the mean BL value for only that cohort of participants with data available at that visit.
Time Frame: BL, Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 212 | 98
units on a scale
  Day 169 cohort (n=212, n=98) | -25.0 (1.95) | -7.28 (2.86)
  Day 365 cohort (n=204, n=97) | -26.1 (2.10) | -21.8 (2.77)
  Day 729 cohort (n=157, n=74) | -28.2 (2.08) | -22.2 (3.71)
  Day 1093 cohort (n=135, n=59) | -28.4 (2.53) | -24.6 (4.58)
  Day 1457 cohort (n=119, n=50) | -26.9 (2.52) | -25.8 (4.60)
  Day 1821 cohort (n=106, n=47) | -26.8 (3.03) | -28.5 (4.71)

81. Secondary Outcome: OL; Mean Time-matched Baseline Activity Limitation Score Over Time For Participants Treated in the OL
Description: Limitations on activities of daily living in the OL period at each study visit were measured by a 2-item questionnaire that was developed to collect data on the amount of time that a participant is unable to perform their usual activities because of their rheumatoid arthritis. Time-matched baseline values were presented by visit and represented the mean baseline value for only that cohort of participants with data available at that visit. The scale ranges from 0 to 100 with increasing score indicating increasing restrictions on levels of activity.
Time Frame: BL
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 206 | 94
units on a scale
  Day 169 cohort (n=206, n=94) | 17.18 (11.09) | 15.01 (11.34)
  Day 365 cohort (n=196, n=93) | 16.97 (11.17) | 15.70 (11.29)
  Day 729 cohort (n=150, n=72) | 16.59 (11.40) | 14.56 (10.87)
  Day 1093 cohort (n=128, n=56) | 15.66 (11.26) | 15.38 (10.94)

82. Secondary Outcome: OL; Mean Change From Baseline in Activity Limitation Score Over Time For Participants Treated in the OL
Description: Limitations on activities of daily living in the OL period at each study visit was measured by a 2-item questionnaire that was developed to collect data on the amount of time that a participant is unable to perform their usual activities because of their rheumatoid arthritis. The scale ranges from 0 to 100 with increasing score indicating increasing restrictions on levels of activity.
Time Frame: Days 169, 365, 729, 1093, 1457, and 1821
Population: as for outcome 8
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OL: ABA | OL: PLA
Number analyzed (Participants) | 206 | 94
units on a scale
  Day 169 cohort (n=206, n=94) | -7.80 (0.83) | -1.78 (1.01)
  Day 365 cohort (n=196, n=93) | -8.04 (0.91) | -6.08 (0.98)
  Day 729 cohort (n=150, n=72) | -8.29 (1.00) | -8.32 (1.25)
  Day 1093 cohort (n=128, n=56) | -8.98 (1.09) | -8.88 (1.51)

83. Secondary Outcome: Cumulative Analysis (DB + OL); Number of Participants With Positive Anti-Abatacept or Anti-Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Responses by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: as for outcome 36
Time Frame: From BL (Day 1) to Day 1821
Population: All participants treated on study with at least one post-baseline immunogenicity measurement.
Measure: Number; unit: participants
Groups:
- All Treated Participants: Participants with active RA who met the inclusion/exclusion criteria for this study were randomized to receive either abatacept or placebo on a background of DMARDs. Participants must have been treated with anti-TNF therapy for at least 3 months and designated as anti-TNF therapy failures due to inadequate efficacy. Participants weighing < 60 kg received 500 mg, participants weighing 60 kg to 100 kg received 750 mg, and participants weighing > 100 kg received 1 gram of abatacept. Abatacept or placebo was administered on Days 1, 15, 29 and every 28 days thereafter for a total of 7 doses. Each dose was infused intravenously over approximately 30 minutes.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 329
participants
  Anti-abatacept antibodies | 22
  Anti-CTLA4 antibodies | 5
  Total | 26

ADVERSE EVENTS:
Groups:
- Open-label ABA: All participants who completed the double-blind period were eligible to continue in the open-label period. At the beginning of the open-label period (Day 169), all eligible participants were re-allocated to a 10 mg/kg weight-tiered dose of abatacept at their enrollment visit into the open-label period. Participants weighing > 100 kg received 1 g, participants weighing ≥ 60 kg and ≤ 100 kg received 750 mg, and participants weighing < 60 kg received 500 mg on a background of DMARDs (at discretion of the investigator). Concomitant biologic RA therapies were later excluded.
Arm/Group | Open-label ABA | Abatacept (ABA) | Placebo (PLA)
Serious Adverse Events (participants affected / at risk) | 136/317 | 28/258 | 16/133
Other Adverse Events (participants affected / at risk) | 276/317 | 153/258 | 65/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label ABA (N=317) | Abatacept (ABA) (N=258) | Placebo (PLA) (N=133)
WEIGHT DECREASED (Investigations) | 1 | 0 | 0
BLOOD GLUCOSE DECREASED (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM CHANGE (Investigations) | 1 | 0 | 0
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 1 | 0 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1 | 0
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 2 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0
HAEMATOMA (Vascular disorders) | 1 | 0 | 0
ISCHAEMIA (Vascular disorders) | 1 | 0 | 0
HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 3 | 1 | 0
PERIPHERAL EMBOLISM (Vascular disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 0
LIVER INJURY (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 5 | 1 | 0
CYTOLYTIC HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 0
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 2 | 0 | 0
AMYLOIDOSIS (Immune system disorders) | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 2 | 0 | 0
DEMENTIA (Nervous system disorders) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 2 | 0 | 0
SCIATICA (Nervous system disorders) | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 1 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0
RADICULOPATHY (Nervous system disorders) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0
NERVE COMPRESSION (Nervous system disorders) | 0 | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
JEJUNITIS (Gastrointestinal disorders) | 1 | 0 | 0
PERITONITIS (Gastrointestinal disorders) | 1 | 0 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 1
HERNIAL EVENTRATION (Gastrointestinal disorders) | 2 | 0 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 2 | 0 | 1
PNEUMONIA (Infections and infestations) | 10 | 1 | 0
PYOTHORAX (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 2 | 0 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 1 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0
RECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0
GRAFT INFECTION (Infections and infestations) | 1 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 5 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
BURSITIS INFECTIVE (Infections and infestations) | 1 | 0 | 0
KERATITIS HERPETIC (Infections and infestations) | 1 | 0 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 1 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 1 | 0
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0 | 0
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0
SUBACUTE ENDOCARDITIS (Infections and infestations) | 1 | 0 | 0
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0
ENTEROBACTER PNEUMONIA (Infections and infestations) | 1 | 0 | 0
PERIORBITAL CELLULITIS (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0
PERIDIVERTICULAR ABSCESS (Infections and infestations) | 0 | 1 | 0
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 3 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 1
CALCULUS URETHRAL (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1 | 0
OBESITY (Metabolism and nutrition disorders) | 3 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
CYSTOCELE (Reproductive system and breast disorders) | 1 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 1 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 1 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 2 | 0 | 1
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 | 0 | 1
UTERINE POLYP (Reproductive system and breast disorders) | 1 | 0 | 0
BREAST ATROPHY (Reproductive system and breast disorders) | 1 | 0 | 0
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0
ADNEXA UTERI MASS (Reproductive system and breast disorders) | 0 | 0 | 1
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 | 0 | 0
URETHRAL INTRINSIC SPHINCTER DEFICIENCY (Congenital, familial and genetic disorders) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0
CORNEAL SCAR (Injury, poisoning and procedural complications) | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 6 | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 2 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 3 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
DEVICE DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
FAILURE OF IMPLANT (Injury, poisoning and procedural complications) | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 0 | 1 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 13 | 2 | 1
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
RHEUMATOID NODULE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 42 | 5 | 3
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SINUS POLYP (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY CAVITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PAIN (General disorders) | 0 | 0 | 2
DEATH (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 6 | 0 | 1
IMPAIRED HEALING (General disorders) | 0 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0 | 0
ADVERSE DRUG REACTION (General disorders) | 1 | 0 | 0
CATHETER SITE HAEMORRHAGE (General disorders) | 1 | 0 | 0
MECHANICAL COMPLICATION OF IMPLANT (General disorders) | 1 | 0 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
THYROID CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label ABA (N=317) | Abatacept (ABA) (N=258) | Placebo (PLA) (N=133)
HYPERTENSION (Vascular disorders) | 43 | 10 | 4
INSOMNIA (Psychiatric disorders) | 21 | 7 | 3
DEPRESSION (Psychiatric disorders) | 24 | 6 | 3
SEASONAL ALLERGY (Immune system disorders) | 18 | 1 | 0
HEADACHE (Nervous system disorders) | 51 | 32 | 7
DIZZINESS (Nervous system disorders) | 33 | 11 | 5
NAUSEA (Gastrointestinal disorders) | 47 | 17 | 8
VOMITING (Gastrointestinal disorders) | 23 | 6 | 3
DIARRHOEA (Gastrointestinal disorders) | 49 | 14 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 17 | 6 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 20 | 4 | 2
INFLUENZA (Infections and infestations) | 32 | 6 | 3
SINUSITIS (Infections and infestations) | 59 | 15 | 5
BRONCHITIS (Infections and infestations) | 66 | 15 | 6
HERPES ZOSTER (Infections and infestations) | 18 | 4 | 3
TOOTH ABSCESS (Infections and infestations) | 18 | 1 | 1
GASTROENTERITIS (Infections and infestations) | 22 | 2 | 1
NASOPHARYNGITIS (Infections and infestations) | 61 | 20 | 8
URINARY TRACT INFECTION (Infections and infestations) | 56 | 7 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 105 | 15 | 10
ANAEMIA (Blood and lymphatic system disorders) | 16 | 3 | 3
RASH (Skin and subcutaneous tissue disorders) | 31 | 6 | 3
FALL (Injury, poisoning and procedural complications) | 23 | 9 | 7
CONTUSION (Injury, poisoning and procedural complications) | 17 | 8 | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 19 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 54 | 15 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 43 | 12 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 1
FATIGUE (General disorders) | 30 | 8 | 6
PYREXIA (General disorders) | 20 | 6 | 2
CHEST PAIN (General disorders) | 23 | 2 | 1
OEDEMA PERIPHERAL (General disorders) | 20 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.